


# **Statistical Analysis Plan**

**BI Study Number 1160-0297** 

Protocol Version 1.0. Date: 24 May 2019

Non-Interventional, cross-sectional study to describe NOACs management in elderly patients with non-valvular atrial fibrillation (NVAF) in Spain. RE-BELD Study

VERSION NUMBER AND DATE: VERSION 1.0; 08 JULY 2020

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx

Author: Version Number: Version 1.0

Version Date: [08072020]

Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




# STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan < Version 1.0, 08 JULY 2020> for Protocol 1160-0297.

| | Name | Signature | Date | |
|---|---|---|---|---|
| Author: | | DocuSigned by: | 10-jul2020 01:55 | 5 PDT |
| Position: | Statistician | Nombre del firmante:<br>Motivo de la firma: Soy el autor de es<br>Hora de firma: 10-jul2020 01:55 Pl | | |
| Company: | | | | |

| | Name | Signature | Date |
|---|---|---|---|
| Approved By: | | DocuSigned by: | 13-jul2020 01:28 F |
| Position: | Project | Nombre del firmante: Motivo de la firma: He revisado este documento Hora de firma: 13-jul2020 01:28 PDT | |
| Company: | | | |
| | | DocuSigned by: | |
| Approved By: | | Signer Name: | 13-Jul-2020 11:05 C |
| Position: | Medical Project | Signing Reason: I approve this document<br>Signing Time: 13-Jul-2020 11:04 CEST | • |
| Company: | | | |
| | | DocuSigned by: | |
| Approved By: | | Signer Name: | 13-Jul-2020 17:36 C |
| Position: | Global Statistician | Signing Reason: I have reviewed this docur<br>Signing Time: 13-Jul-2020 17:36 CEST | ment |
| Company: | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 05Jan2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




# **MODIFICATION HISTORY**

| Unique | Date of the | Author | Significant Changes from |
|-------------|--------------|--------|------------------------------|
| Identifier | Document | | Previous Authorized Version |
| for this | Version | | |
| Version | | | |
| Draft 1.0 | 29-OCT-2019 | | Not Applicable – First draft |
| Draft 2.0 | 28-FEB-2020 | _ | No |
| Draft 3.0 | 22-MAY-2020 | | No |
| Draft 4.0 | 05-JUNE-2020 | | No |
| Draft 5.0 | 25-JUNE-2020 | | No |
| Draft 6.0 | 08-JULY-2020 | | No |
| Version 1.0 | 08-JULY-2020 | | No |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




Reference: RWI\_WI\_BIOS0015

# **TABLE OF CONTENTS**

| 1. | ABB | REVIATI | IONS | 7 |
|---|---|---|---|---|
| <b>2.</b> | INTE | RODUCT | ION | 9 |
| <b>3.</b> | STU | DY OBJE | CCTIVES | 9 |
| | 3.1 | Primary | Objectives | 9 |
| | 3.2 | Seconda | ary Objectives | 9 |
| 4. | STU | DY DESI | ĠŇ | 10 |
| | 4.1 | General | Description | 10 |
| | 4.2 | | ize | |
| | 4.3 | • | tion of treatment | |
| | 4.4 | Study fl | low/schedule | 13 |
| | 4.5 | Schedul | le of Events | 14 |
| | 4.6 | Change | s to Analysis from Protocol | 14 |
| <b>5.</b> | PLA] | | NALYSES | |
| | 5.1 | | Analysis | |
| | 5.2 | Final A | nalysis | 15 |
| <b>6.</b> | ANA | LYSIS SI | ETS | 15 |
| | 6.1 | All Sub | jects Enrolled Set [ENR] | 15 |
| | 6.2 | Full An | alysis Set [FAS] | 15 |
| | 6.3 | Safety A | Analysis Set [SAF] | 16 |
| <b>7.</b> | GEN | ERAL C | ONSIDERATIONS | 16 |
| | 7.1 | Referen | ce Start/End Date | 17 |
| | 7.2 | Commo | on Calculations | 18 |
| | | 7.2.1 | Weight | 18 |
| | | 7.2.2 | Body Mass Index (BMI) | 18 |
| | | 7.2.3 | Charlson Comorbidity Index | |
| | | 7.2.4 | Laboratory values | 20 |
| | | 7.2.5 | Time since NVAF diagnosis | 21 |
| | | 7.2.6 | Duration of VKA treatment | 21 |
| | | 7.2.7 | Duration since the first NOAC | 22 |
| | | 7.2.8 | Duration since NVAF diagnosis until first NOAC | |
| | | | initiation | 22 |
| Dod | cument: | | R-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto | o\Estadistica\SAP\S |
| Aut | hor: | AP_REE | BELD_version1.0_08072020.docx Version Number: | Version 1.0 |

Effective Date: 15Jun2018

Template No.: RWI\_TP\_BIOS0013 Revision 1

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




Reference: RWI\_WI\_BIOS0015

| | | 7.00 | D CC DIOLG | | 22 |
|---|---|---|---|---|---|
| | | 7.2.9 | | nent | |
| | | 7.2.10 | | nents | |
| | | 7.2.11 | | | |
| | | 7.2.12 | | | |
| | | 7.2.13 | | ntiplatelet agents | |
| | | 7.2.14 | | | |
| | | 7.2.15 | | | |
| | | 7.2.16 | | | 25 |
| | | 7.2.17 | Underdosed or overdosed patie treatment) | ent (current NOAC | 25 |
| | 7.3 | Software | Version | | |
| 8. | | | CONSIDERATIONS | | |
| | 8.1 | | l Bias Reduction | | |
| | 8.2 | | l Tests and Confidence Intervals | | |
| | 8.3 | | ents for Covariates and Factors to | | |
| | 8.4 | | data | | |
| | 8.5 | | tion of Subgroups | | |
| 9. | | PHT PRES | SENTATIONS | | 29 |
| ).<br>10. | | | AND WITHDRAWALS | | |
| 10.<br>11. | | | IC AND OTHER BASELINE | | |
| 11. | 11.1 | | ons | | |
| 12. | | | S. | | |
| 13. | | | CATION EXPOSURE | | |
| 13.<br>14. | | | | | |
| 17. | 14.1 | | Outcome | | |
| | 17.1 | 14.1.1 | | Outcome | |
| | 14.2 | | ry Outcomes | | |
| | 17.2 | 14.2.1 | | | |
| | | 14.2.2 | | | |
| | | 14.2.3 | | | |
| | | 14.2.4 | | | |
| | 14.3 | | of Secondary Outcomes | | |
| | 14.3 | • | • | | |
| | | 14.3.1<br>14.3.2 | | | |
| | | 14.3.3 | <u> </u> | | |
| Doc | ument: | | Europe\2019\2512352 - Study on anticoagu<br>ELD_version1.0_08072020.docx | ilation management - BI\Proyecto\Estadist | tica\SAP\S |
| Autl | nor: | Ar_nebe | LLD_VEISIONIT.U_U0U72U2U.UUCX | Version Number: | Version 1.0 |
| | | | | version bate. | [000/2020] |

Effective Date: 15Jun2018

Template No.: RWI\_TP\_BIOS0013 Revision 1

and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




| | | 14.3.4 | Prevention strategy | 36 |
|---|---|---|---|---|
| | 14.6 | Explorat | tory analysis | 38 |
| 15. | SAFE | | | |
| | 15.1 | Adverse | Drug Reactions | 39 |
| | 15.2 | | Adverse Drug Reactions | |
| | 15.3 | | | |
| 16. | REFE | | S | |
| <b>17.</b> | | | MOCK TABLES | |
| | 17.1 | | ty | |
| | 17.2 | _ | s characteristics | |
| | | 17.2.1 | Patient's characteristics according to current NOAC type | 43 |
| | | 17.2.2 | Patient's characteristics according to duration since the | |
| | | | first NOAC initiation | 62 |
| | 17.3 | Outcome | es | |
| | | 17.3.1 | Primary outcome: Current NOAC | |
| | | 17.3.2 | Secondary outcome: OAC treatment management | |
| | | 17.3.3 | Secondary outcome: Clinical Frailty Scale | |
| | | 17.3.4 | Secondary outcome: Prevention strategy | |
| | | 171511 | sociality careement in tention strategy | |
| | 17.4 | Addition | nal tables | 95 |
| | 17.5 | | Drug Reactions | |
| | 17.6 | | Adverse Drug Reactions | |
| | 17.7 | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

 $AP\_REBELD\_version 1.0\_08072020. docx$ 


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




### 1. ABBREVIATIONS

ACE Angiotensin Converting Enzyme inhibitors

ADR Adverse Drug Reaction
AF Atrial Fibrillation

AIDs Acquired immune deficiency syndrome

ALT Alanine Aminotransferase
ARB Angiotensin-Receptor Blockers
AST Aspartate Aminotransferase
BI Boehringer Ingelheim

BID Twice a day
BMI Body Mass Index

CABG Coronary Artery Bypass Grafting CCI Charlson Comorbidity Index

CFS Clinical Frailty Scale

CHA2DS2-VASc Congestive heart failure, Hypertension, Age (> 75), Diabetes mellitus,

Stroke/TIA, Vascular disease, Age 65-74, Sex Category

CI Confidence Interval
CKD Chronic Kidney Disease
CRF Case Report Form

eCRF Electronic Case Report Form

EHRA European Heart Rhythm Association

GFR Glomerular Filtration Rate

HAS-BLED Hypertension, Abnormal renal and liver function, Stroke (1 point),

Bleeding history or predisposition, Labile INR, Elderly (>65 years),

Drugs and Alcohol.

ICH Intracranial haemorrhage

ICH-GCP Harmonized Tripartite Guideline for Good Clinical Practice

INR International Normalized Ratio
LVEF Left ventricular ejection fraction
NSAIDs Nonsteroidal Anti-Inflammatory Drugs

NYHA New York Heart Association

NOAC Non-vitamin K antagonist oral anticoagulant

NVAF Non-valvular atrial fibrillation

OAC Oral anticoagulant

PCI Percutaneous coronary intervention

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP REBELD version1.0 08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




PT Preferred Terms
QD Once a day

SADR Serious Adverse Drug Reaction SAHS Sleep apnoea-hypopnoea syndrome

SAP Statistical Analysis Plan

SmPC Summary of Product Characteristics

SOC System Organ Classes

SOPs Standard Operating Procedures
TIA Transitory ischemic attack
TLF Tables/Listings/Figures
VKA Vitamin K Antagonist

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




#### 2. INTRODUCTION

This statistical analysis plan (SAP) describes the rules and conventions to be used in the presentation and analysis of treatment patterns and patient profile. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed. This statistical analysis plan (SAP) is based on protocol version 1.0, dated 24 May 2019 and case report forms (CRFs) version 2, dated 10 March 2020.

#### 3. STUDY OBJECTIVES

This study has been designed in order to describe the current non-vitamin K antagonist oral anticoagulants (NOACs) management in elderly patients in Spain.

# 3.1 Primary Objectives

The primary objective is to describe the pattern of usage of NOACs prescribed according to their Summary of Product Characteristics (SmPC), by current NOAC type and dose, in elderly patients (≥75 years-old) with non-valvular atrial fibrillation (NVAF) at the time of the study visit.

# 3.2 Secondary Objectives

The secondary objectives are:

- 1. To describe patients' characteristics at the time of the study visit by current NOAC type stratified by duration since first NOAC initiation.
- 2. To describe OAC treatment management since first NOAC initiation until the study visit by duration since first NOAC initiation: previous vitamin K antagonists (VKA) treatment, first NOAC treatment duration, dose changes, switch between NOACs and

Document:

 $\label{lem:hamman} \mbox{H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\SAP\SAP\ABOR_Europe\ABOR_Eur$ 

AP\_REBELD\_version1.0\_08072020.docx

Author:

Version Number:

Version 1.0

Version Date:

[08072020]

Template No.: RWI TP BIOS0013 Revision 1

Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




reasons for switch, total NOAC treatment duration and additional antiplatelet treatment.

- 3. To describe the Clinical Frailty Scale grading, CFS (1), at the time of the study visit, by current NOAC type.
- 4. To describe first NOAC usage by NOAC type, for primary prevention or secondary prevention, at the time of first NOAC initiation.

**Further objective:** To evaluate the appropriateness of prescribed therapy based on Spanish health authorities' recommendations (2) (therapeutic positioning report) and other regional guidelines by NOAC type (if there are enough patients for a NOAC type), at the time of first NOAC initiation.

#### 4. STUDY DESIGN

# 4.1 General Description

This is an observational, multicenter and cross-sectional study in NVAF elderly patients currently on NOAC treatment for their stroke prevention.

AF is classified as non-valvular AF in the absence of mitral stenosis or cardiac valvular prosthesis, since NOACs are not recommended for patients with mechanical heart valve (level of evidence B) or moderate to severe mitral stenosis (level of evidence C) (3).

The study will be conducted in approximately 50 sites in Spain. Investigators from different specialties are planned to be included as follows: 35 cardiologists, 10 hematologists and 5 geriatricians.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP REBELD version1.0 08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




The design of the study imposes a single visit to be performed for the informed consent signature and data collection that will coincide with one of those performed by the patients as part of routine follow-up of their disease, without interfering with usual clinical practice of the investigator.

A specific therapeutic strategy has already been assigned to each included patient, based on routine practice and without interference with the physician's prescription habits. The observational nature of the study is ensured as no diagnostic or therapeutic intervention outside of routine clinical practice will be applied.

Cardiology, hematology, geriatric services at a hospital setting, specialty medical offices and nursing homes, who regularly prescribe NOACs for stroke prevention in NVAF patients may be invited to participate.

The number of patients per site to be included in the study will be initially set up to a maximum of 10 patients per site. Once the 50% of the participating sites have been initiated, the recruitment will become competitive until the end of the study and the limitation of 10 patients per site will be removed to allow sites to continue with the recruitment.

# 4.2 Study size

It is planned that a total of approximately 500 patients will be recruited for the study. Based on such a sample size estimate, categorical variables of binomial proportions (e.g. sex) will be estimated with the precision (i.e. width of descriptive 95% confidence interval) described in the following Table 1. Calculations of the confidence intervals (CI) are based on the Clopper-Pearson method:

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to


Table 1. Width of 95% confidence interval by prevalence

| Prevalence of attribute | Sample size |
|-------------------------|-------------|
| | 500 |
| 10% Expected n | 50 |
| 95% CI width | 5.46% |
| 20% Expected n | 100 |
| 95% CI width | 7.20% |
| 30% Expected n | 150 |
| 95% CI width | 8.22% |
| 40% Expected n | 200 |
| 95% CI width | 8.76% |
| 50% Expected n | 250 |
| 95% CI width | 8.76% |

# 4.3 Description of treatment

Patients in this study will be currently on treatment with NOAC for their NVAF, according to the indication approved in their SmPC, and initiated it at least 3 months before the study visit. Prescription of the treatments will have been done under the sole responsibility of the healthcare professional and before considering the participation in the study.

In addition, no intervention, either diagnostic or therapeutic, will be applied to patients other than that used for routine clinical practice.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018




# 4.4 Study flow/schedule

The design of the study imposes a single visit to be performed for the informed consent signature and data collection that will coincide with one of those performed by the patients as part of routine follow-up of their disease, without interfering with usual clinical practice of the investigator.

Figure 1. Study scheme for study period



After signing the informed consent, investigator will assess the Clinical Frailty Scale (1), the Modified EHRA scale for AF related symptoms (4), the NYHA classification of heart failure (5) and the CHA2DS2-VASc and HAS-BLED scales and include the scores directly in eCRF after evaluating the patient's functional status and patient's medical records. The investigator will review the medical records in order to complete other variables needed to address study objectives that will mainly be obtained directly from patient medical records or requested to the patient at the study visit if not available in medical records. The end of the single study visit is the end of the study for each patient.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




#### 4.5 Schedule of Events

The schedule of events can be found in Section 6 of the protocol (Milestones).

# 4.6 Changes to Analysis from Protocol

Per protocol, the variable "reason for VKA switch will be described under the OAC treatment management outcome. Finally, reason for VKA treatment switch has not been collected specifically in the VKA section of the CRF. This has been deleted from section 14.2.2 of SAP.

New analysis not included in the final protocol have been considered:

- Antiplatelet treatment according to current NOAC type
- Treatment received at the moment of thromboembolic and bleeding events.
- For all NOACs, the different doses that patients take according to HAS-BLED score.
- Underdosed and overdosed patients (for current NOAC treatment).
- HAS-BLED total score according to NOAC and antiplatelet current treatment.
- Multivariate model to evaluate the association between the Clinical Frailty Scale (dependent variable) and the thromboembolic and the bleeding events (independent variables). To calculate this analysis, only events that have occurred subsequent to the start of anticoagulant therapy (not those prior to the start of VKA / NOACs) will be considered. Univariate analysis will be performed. All variables which have a P value of less than 0.1 will be included in the multivariate analysis.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018




#### 5. PLANNED ANALYSES

#### 5.1 **Interim Analysis**

No interim analysis has been planned.

#### 5.2 **Final Analysis**

All final, planned analyses identified in this SAP will be performed by Real-World Evidence Solutions (RWES) Biostatistics following SOPs. Final CSR will be performed using Boehringer Ingelheim template.

#### 6. **ANALYSIS SETS**

#### 6.1 All Subjects Enrolled Set [ENR]

The all subjects enrolled (ENR) set will contain all subjects who provide informed consent for this study.

#### 6.2 **Full Analysis Set [FAS]**

The full analysis set (FAS) will contain all enrolled subjects who provide informed consent for this study (ENR set) and fulfill all selection criteria. This is called "eligible patients" in the protocol.

Patients will be included in FAS if all of the following criteria are met:

- 1. Patients are willing and provide written informed consent prior to participate in this study
- 2. Patients  $\geq$  75 years-old at the time of the study visit.
- 3. Patients with a diagnosis of non-valvular atrial fibrillation (NVAF).

H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S Document: AP\_REBELD\_version1.0\_08072020.docx Author: Version Number: Version 1.0 [08072020] Version Date:

Reference: RWI WI BIOS0015 Template No.: RWI TP BIOS0013 Revision 1

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




- 4. Patients who are being treated with NOAC treatment according to the indication approved in the SmPC.
- 5. Patients who have started the NOAC treatment at least 3 months prior to the study visit.

Patients will be excluded from participating in this study, and will be excluded from this analysis set, if the following criterion is met:

- 1. Current participation in any clinical trial of a drug or device.
- 2. Patients who have any contraindication for NOAC treatment, according to the SmPC.

# 6.3 Safety Analysis Set [SAF]

The safety analysis set (SAF) will contain all enrolled subjects who receive at least one documented dose of Pradaxa®.

#### 7. GENERAL CONSIDERATIONS

The design of the study imposes a single visit to be performed and that will coincide with one of those performed by the patients as part of routine follow-up of their disease, without interfering with usual clinical practice of the investigator.

Data will be collected through an eCRF which will include all the study variables. Investigator will enter patient data in eCRF. Variables collected at the time of the study visit (including those related to the first NOAC initiation) will be obtained based on and limited to those available in the medical records of the selected patients. Demographic characteristics, smoking habit and alcohol consumption may be asked to the patient at the study visit if not available in the medical records. LVEF measurement will be obtained from the last images available for the patient.

Document:

 $\label{thm:hamman} \mbox{H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\SAP\SAP\ABOR_Europe\ABOR_Eur$ 

AP REBELD version1.0 08072020.docx

Author:

Version Number: Version 1.0


Template No.: RWI\_TP\_BIOS0013 Revision 1

Reference: RWI WI BIOS0015

Effective Date: 15Jun2018




Clinical Frailty Scale, modified EHRA scale for AF related symptoms, NYHA classification for heart failure, CHA2DS2-VASc and HAS-BLED scores will be assessed by the investigators at the study visit by evaluating the patient's functional status and medical records and the values will be directly included in the eCRF.

Final score for the Comorbidities Charlson Index will be automatically calculated based on the answers individually entered by the investigator in the eCRF for each index item (6).

Any required missing data to calculate the score for the scales or the Comorbidities Charlson Index may be asked to the patient at the study visit if not available in the medical records and should be documented, however the final score number obtained by the investigator from this information will not need to be included in medical records.

Boehringer Ingelheim reserves the right to discontinue the study overall or at a particular study site at any time for the following reasons:

- 1. Failure to meet expected enrolment goals overall or at a particular study site
- 2. Administrative reasons (i.e. study rejected by the hospital director)
- 3. Violation of GxP (as applicable), the study protocol, or the contract by a study site or investigator, disturbing the appropriate conduct of the study

#### 7.1 Reference Start/End Date

Reference start date is date of study visit, collected in the eCRF as a mandatory variable.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




# 7.2 Common Calculations

### **7.2.1** Weight

Weight (kg) will be categorized in two categories according to dose adjustment criteria in NOAC:

- ≤60 kg
- >60 kg

# 7.2.2 Body Mass Index (BMI)

The formula to obtain Body Mass Index is the following: BMI (kg/ m²) = weight (kg)/ height² (m) and BMI will be categorized into 5 categories according to the World Health Organization (WHO):

- Underweight: BMI< 18.5 kg/m<sup>2</sup>
- Normal weight:  $18.5 \text{ kg m}^2 \le BMI \le 25 \text{ kg/m}^2$
- Overweight:  $25 \text{ kg/m}^2 < \text{BMI} <= 30 \text{ kg/m}^2$
- Obese:  $30 \text{ kg/m}^2 < BMI <= 35 \text{ kg/m}^2$
- Severely Obese: BMI> 35 kg/m<sup>2</sup>

#### 7.2.3 Charlson Comorbidity Index

The Charlson Comorbidity Index (CCI) predicts the ten-year mortality for patients presenting one or more of the conditions in the model, where the age groups and each condition are awarded a specific number of points, some conditions weighing more than others, based on the adjusted risk of mortality. The more points given, the more likely the predicted adverse outcome. The index then sums the points and offers a 10-year survival/ mortality prognosis.

https://www.thecalculator.co/health/Charlson-Comorbidity-Index-(CCI)-Calculator-765.html https://www.mdcalc.com/charlson-comorbidity-index-cci

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018




Each of the conditions listed below are awarded 1, 2, 3 or 6 points depending on the mortality risk. CCI will be calculated as the sum of all points included in the following table:

Table 2. Point assigned to Charlson Comorbidity Index

| | POINTS |
|-------------------------------------------------------|--------|
| Age | |
| 50–59 years | +1 |
| 60–69 years | +2 |
| 70–79 years | +3 |
| >=80 years | +4 |
| Myocardial infarction | +1 |
| Congestive Heart Failure (CHF) | +1 |
| Peripheral vascular disease | +1 |
| Cerebrovascular Accident or Transient ischemic attack | +1 |
| COPD | +1 |
| Connective tissue disease | +1 |
| Peptic ulcer disease | +1 |
| Liver disease | |
| Mild | +1 |
| Moderate to severe | +3 |
| Diabetes mellitus | |
| Uncomplicated | +1 |
| End-organ damage | +2 |
| Hemiplegia | +2 |
| Moderate to severe* Chronic Kidney Disease (CKD) | +2 |
| Solid tumor | |
| Localized | +2 |
| Metastatic | +6 |
| Leukemia | +2 |
| Lymphoma | +2 |
| AIDS | +6 |

Document:

 $\label{thm:hor-europe} \end{\colored} H:\hor-Europe\colored anticoagulation management-BI\proyecto\Estadistica\SAP\Sample\Samp$ 

AP\_REBELD\_version1.0\_08072020.docx

Author:


Template No.: RWI TP BIOS0013 Revision 1

Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

<sup>.</sup> and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




# 7.2.4 Laboratory values

#### 7.2.4.1 Serum creatinine

Serum creatinine will be categorized in two categories (7):

- Normal levels: 0.6-1.2 mg/dl in males and 0.5-1.1 mg/dl in females
- High/low levels

#### 7.2.4.2 Creatinine clearance

Creatinine clearance will be estimated using Cockcroft-Gault formula (7):

 $CCr = (140 - Age(years)) \times Weight(kg) \times [0.85 \text{ if female}] / 72 \times [Serum Creatinine (mg/dL)]$ 

Chronic Kidney Disease will be categorized according to these values, included in Clinical Practice Guidelines for Chronic Kidney Disease: Evaluation, Classification, and Stratification:

- $\geq$ 90: Kidney damage with normal or increased glomerular filtration rate (GFR)
- 60-89: Kidney damage with mild decreased GFR
- 30-59: Moderate decrease in GFR
- 15-29: Severe decrease in GFR
- <15: Kidney failure

#### 7.2.4.3 ALT, AST and bilirubin values

ALT, AST and bilirubin will be categorized in two categories, according to (https://www.org/tests-procedures/liver-function-tests/about/pac-20394595):

# ALT (GPT):

- Normal values: 7-55 UI/L
- High/low values

# AST (GOT):

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




- Normal values: 8-48 UI/L
- High/low values

#### Bilirubin:

- Normal values: 0.2-1.2 mg/dl
- High/low values

# 7.2.4.4 Haemoglobin and platelets

Haemoglobin and platelets levels will be categorized in two categories, according to American cancer society (<a href="https://www.cancer.org/content/dam/CRC/PDF/Public/7174.pdf">https://www.cancer.org/content/dam/CRC/PDF/Public/7174.pdf</a>):

- Normal values: 12-18 g/dL
- High/low values

#### Platelets:

Haemoglobin:

- Normal values: 150-450 x103/μL
- High/low values

# 7.2.5 Time since NVAF diagnosis

The number of years since diagnosis will be obtained from number of years between date of NVAF diagnosis and date of study visit as follows:

Time of NVAF evolution (years) = (date of study visit – date of NVAF diagnosis + 1)/(365.25).

#### 7.2.6 **Duration of VKA treatment**

VKA treatment duration in years will be calculated as number of months/12 (in case of months specified). In case of more than one VKA treatment, the total VKA treatment duration will be calculated as the sum of the years in treatment of each one.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018




#### 7.2.7 Duration since the first NOAC

The number of months since the first NOAC initiation date until the study visit date will be obtained as follows:

Duration since the first NOAC (months) = (date of study visit – date of first NOAC + 1)/(30.5). Duration since the first NOAC initiation until study visit will be categorized as >4 months and <4 months.

#### 7.2.8 Duration since NVAF diagnosis until first NOAC initiation

The number of months since the NVAF diagnosis date until the first NOAC initiation date will be obtained as follows:

Duration since the NVAF diagnosis until first NOAC initiation (months) = (date of first NOAC – date of NVAF diagnosis + 1)/(30.5).

#### 7.2.9 Duration of first NOAC treatment

The duration of the first NOAC treatment will be calculated as the number of years (or months, depending on the data) between stop date and start date for the NOAC treatment with the minimum start date:

Duration of the first NOAC (years) = (stop date of first NOAC – start date of first NOAC + 1)/(365.25) or

Duration of the first NOAC (months) = (stop date of first NOAC – start date of first NOAC + 1)/(30.5)

In the case the first NOAC has not been finished, the study visit date will be considered as the stop date (censured cases).

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




#### 7.2.10 Duration of new NOAC treatments

The duration of new NOAC treatment will be calculated as the number of years (or months, depending on the data) between stop date and start date for the new NOAC treatment:

Duration of the new NOAC (years) = (stop date of new NOAC – start date of new NOAC + 1)/(365.25). or

Duration of the new NOAC (months) = (stop date of new NOAC – start date of new NOAC + 1)/(30.5).

In the case the new NOAC has not been finished, the study visit date will be considered as the stop date.

#### 7.2.11 Total time in NOAC treatment

NOAC treatment duration in years will be calculated as the sum of the years of each NOAC treatment. The duration of the each NOAC treatment will be calculated as:

Duration of each NOAC (years) = (stop date of NOAC – start date of NOAC + 1)/(365.25).

For the last NOAC treatment (receiving at study visit) the stop date will be the study visit date.

In other hand, in the case there are periods of interruption of the NOAC treatment, only the time that they have been in treatment will be considered. In this case, the time in each period will be calculated from the previous formula, adding the different periods in treatment.

#### 7.2.12 Number of switches

The number of switches will be defined as the number of changes to another NOAC.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




# 7.2.13 Total time in treatment with antiplatelet agents

Time in treatment with antiplatelet agents (in years or months) will be calculated as the sum of the years of each antiplatelet treatment. The duration of each antiplatelet treatment will be calculated as:

Duration of the each antiplatelet (years) = (stop date of antiplatelet – start date of antiplatelet + 1)/(365.25).

Duration of the each antiplatelet (months) = (stop date of antiplatelet – start date of antiplatelet + 1)/(30.5).

For the last antiplatelet treatment (if it is received at study visit) the stop date will be the study visit date.

# 7.2.14 Clinical Frailty Scale (CFS)

The CFS score will be categorized in two categories, according to this ranges:

- 1) Frailty patients CFS scoring >4
- 2) Non-frailty patients CFS scoring ≤4

#### 7.2.15 CHA2DS2-VASc Scale

The CHA2DS2-VASc total score will be categorized in three categories, according to the risk of stroke (8):

- 1) Low risk (score 0 in male; score 1 in female)
- 2) Moderate risk (score 1 in male; score 2 in female)
- 3) High risk (score  $\geq 2$  in male; score  $\geq 3$  in female)

Note: In the last update of European Society of Cardiology (ESC) guidelines 2016 the "female gender" is no longer considered by itself as an increase of the risk.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




#### 7.2.16 HAS-BLED Scale

The HAS-BLED total score will be categorized in three categories, according to the bleeding risk (9):

- 1) Low risk (score 0)
- 2) Intermediate risk (score 1-2)
- 3) High risk (score  $\geq$ 3)

# 7.2.17 Underdosed or overdosed patient (current NOAC treatment)

The recommended dose of dabigatran is 150mg twice a day (BID). Patients who meet any of the following criteria should perform a dose adjustment to 110mg BID, so those who receive the recommended dose of 150mg BID will be classified as overdosed. Those who receive a 110mg BID dose and do not meet any of the following criteria will be classified as underdosed:

- Age  $\geq$ 80 years
- Patients aged 75-79 years and HAS-BLED  $\geq$  3
- Moderate renal impairment (creatinine clearance 30-50mL/min)

The recommended dose of rivaroxaban is 20mg once a day (QD). Patients who meet the following criteria should perform a dose adjustment to 15mg QD, so those who receive the recommended dose of 20mg QD will be classified as overdosed. Those who receive a 15mg QD dose and do not meet following criteria will be classified as underdosed:

- Moderate renal impairment (creatinine clearance 30-50mL/min) or severe renal impairment (creatinine clearance 15-29mL/min)

The recommended dose of apixaban is 5mg BID. Patients who meet at least 2 of the following 3 criteria should perform a dose adjustment to 2.5mg BID, so those who receive the

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP REBELD version1.0 08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




recommended dose of 5mg BID will be classified as overdosed. Those who receive a 2.5mg BID dose and do not meet at least 2 of the 3 following criteria will be classified as underdosed:

- Age  $\geq$ 80 years
- Body weight  $\leq 60 \text{ kg}$
- Serum creatinine ≥ 1,5 mg/dl or severe renal impairment (creatinine clearance 15-29mL/min)

The recommended dose of edoxaban is 60mg OD. Patients who meet at least 1 of the following 2 criteria should perform a dose adjustment to 30mg OD, so those who receive the recommended dose of 60mg OD will be classified as overdosed. Those who receive a 30mg OD dose and do not meet at least 1 of the 2 following criteria will be classified as underdosed:

- Body weight  $\leq 60 \text{ kg}$
- Moderate or severe renal impairment (creatinine clearance 15-50mL/min)

A categorical variable for dose category with 3 levels will be described:

- 1) Appropriately dosed
- 2) Underdosed
- 3) Overdosed.

# 7.3 Software Version

All analyses will be conducted using SAS Enterprise Guide version 7.15.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




#### 8. STATISTICAL CONSIDERATIONS

Continuous variables will be described by the number of patients with valid/missing observations, mean, SD, median, 25 and 75 percentiles (Q1 and Q3, respectively), minimum and maximum and categorical variables will be described by frequencies and related percentages. Appendix 1 on page 42 shows the summary TLFs to be provided in the report of the study.

#### 8.1 Statistical Bias Reduction

No statistical methods for handling bias will be used. Given the real-world nature of the data and the descriptive purposes of the study objectives no confounding factor have been identified.

Missing values and drop-outs will be counted in all description of variables, but no imputation will be considered.

#### 8.2 Statistical Tests and Confidence Intervals

No statistical test will be performed.

# 8.3 Adjustments for Covariates and Factors to be Included in Analyses

No statistical modelling will be done. So, no adjustment for covariates and factors to be accounted for in the analyses are considered.

# 8.4 Missing data

Given the real-world nature of the data and the descriptive purposes of most of the study objectives, study variables will not be imputed. Missing values and drop-outs will be counted

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




in all description of variables, but no imputation will be considered. Only date data where the exact day is missing will be imputed, being replaced by the middle of the month.

# 8.5 Examination of Subgroups

Subgroup analyses will be conducted as stated in the exploratory analysis sections. It should be noted that the study was not designed to detect treatment differences within subgroups. The following subgroups will be assessed and described within the exploratory analysis sections (a minimum of 50 patients will be required for each subgroups).

For the primary objective (the pattern of NOAC usage):

- Sex:
  - o Female
  - o Male
- Age at the time of the study visit:
  - o 75-79 years
  - o 80-84 years
  - $\circ$   $\geq$ 85 years
- Presence of each comorbidities at the time of the study visit (heart failure, coronary artery disease, peripheral vascular disease diabetes, chronic kidney disease, liver disease, cancer):
  - o No
  - o Yes

For the secondary objectives (Patient's characteristics at the time of the study visit and OAC treatment management):

• Duration since the first NOAC initiation date until the study visit:

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




- o ≤4 months
- $\circ$  > 4 months

### 9. OUTPUT PRESENTATIONS

Tables and Figures on page 42 describe the presentations for this study and therefore the format and content of the summary TLFs to be provided by

# 10. DISPOSITION AND WITHDRAWALS

All subjects who provide informed consent will be accounted for in this study. Subject disposition, withdrawals, and protocol violations (as defined in section 6.2), including inclusion and exclusion criteria will be presented for all enrolled patients.

# 11. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic data and other baseline characteristics will be presented for the FAS.

The following demographic and other baseline characteristics, related to secondary outcome, will be collected from medical records or at study visit to describe the patient's

characteristics:

Table 3. Patient characteristics at the time of study visit

| | Obtained from | |
|---|---|---|
| | medical | Obtained at the |
| Variable | records | study visit |
| Demographic characteristics: Age, sex, height, weight, BMI, caregiver (Yes/No), place where patient is living (Home alone; At home with | X | X |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| Variable partner/other family member/a friend; Other's home (e.g family member's); Nursing home) | Obtained<br>from<br>medical<br>records | Obtained at the study visit |
|---|---|---|
| Smoking habit (past/current/non-smoker) and alcohol consumption (casual or non-consumer/habitual/abuse/dependence) | Х | x |
| Analytical lab results (from last available blood sample analysis): - Kidney function: serum creatinine (mg/dl), creatinine clearance (Cockcroft-Gault calculation) - Liver function: AST/ALT (UI/L), total bilirubin (mg/dl) - Haemoglobin (g/dl) and platelet levels (x uL) | х | |
| NVAF: - Diagnosis date (month and year) - Type (persistent, long standing persistent, permanent, paroxysmal) - Modified EHRA scale for AF related symptoms | x | x (mEHRA scale) |
| Procedures and interventions: - Cardioversion/Ablation (Yes/No) - Coronary interventions (Yes/No): Percutaneous coronary intervention (PCI)/Coronary Artery Bypass Grafting (CABG) - Pacemaker carrier (Yes/No) | х | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

 $AP\_REBELD\_version 1.0\_08072020. docx$ 


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| Variable | Obtained from medical records | Obtained at the study visit |
|---|---|---|
| Comorbidities and Clinical Risk Factors: - Heart Failure (Yes/No, New York Heart Association (NYHA) classification; Left Ventricular Ejection Fraction, LVEF, %) - Coronary artery disease (Yes/No) - Sleep apnoea-hypopnoea syndrome (SAHS) (Yes/No) - Hypertension (Yes/No) - Hyperlipidemia (Yes/No) - Comorbidity Charlson index (Yes/No; total score): myocardial infarction (already collected for history of thromboembolic events), congestive heart failure (already collected for the NHYA scale scoring), cerebral and peripheral vascular disease, dementia, chronic obstructive pulmonary disease, connective tissue disease, peptic ulcer disease, mild/moderate/severe liver disease, diabetes, diabetes with end-organ damage, hemiplegia, moderate/severe renal disease, any solid tumor, metastatic solid tumor, leukemia, lymphoma AIDs, age (already collected as a demographic characteristic). -History of thromboembolic events (Yes/No, number and date): TIA, ischemic stroke, hemorrhagic stroke, embolism systemic, deep vein thrombosis, pulmonary embolism, stable angina, unstable angina, myocardial infarction with/without ST segment elevation; and bleeding events (Yes/No, number and date): intracranial, digestive, genitourinary, gingival, nasal, pulmonary, articular-muscular, conjunctival. | X | x (NYHA<br>classification,<br>Charlson Index) |
| CHA2DS2-VASc (total score) | | X |
| HAS-BLED (total score) | | X |
| Clinical Frailty Scale | | X |
| Previous vitamin K antagonist (VKA) treatment (yes/no), type | | |
| (acenocoumarol or warfarin), start date and treatment duration Other concomitant treatments (Total number of current concomitant drugs; Type (Yes/No, number): ARB or ACE inhibitor, Beta-blocker, Calcium channel blockers, Diuretics, Amiodarone, Statin, Proton pump inhibitor, H2-receptor antagonist, Digoxin, NSAIDs, Dronedarone, Other antiarrhythmics, ketoconazole (systemic), cyclosporine, itraconazole | х | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




#### 11.1 Derivations

Derived variables are specified in section 7.2 Common Calculations on page 18 in this SAP.

#### 12. MEDICATIONS

Medications will be presented for FAS. In the case of previous treatment with VKA, type, treatment duration will be presented.

Other concomitant treatments in the study visit (ARB or ACE inhibitor, Beta-blocker, Calcium channel blockers, Diuretics, Amiodarone, Statin, Proton pump inhibitor, H2-receptor antagonist, Digoxin, NSAIDs, Dronedarone, Other antiarrhythmics, ketoconazole (systemic), cyclosporine, itraconazole) will be presented.

History and current antiplatelet treatment will be described.

#### 13. STUDY MEDICATION EXPOSURE

Patients in this study will have been prescribed a NOAC treatment for their NVAF. Prescription of the treatments will have been done under the sole responsibility of the healthcare professional and before considering the participation in the study.

#### 14. OUTCOMES

# 14.1 Primary Outcome

The primary outcome is the pattern of usage of non-vitamin K oral anticoagulants (NOACs) prescribed according to their Summary of Product Characteristics (SmPC), based on the percentage of patients by NOAC type and dose the patient is taking at the time of the study visit. Timeframe to complete data collection for this outcome is one day, the study visit day.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018




Table 4. Primary variable collected at the time of the study visit

| Variable | Obtained from medical records |
|----------------------------------------|-------------------------------|
| Current NOAC active substance and dose | X |

### 14.1.1 Primary Analysis of Primary Outcome

The primary outcome analysis will be performed for the FAS. For the primary objective, the pattern of usage of NOAC will be described as the percentage of patients by NOAC type and dose.

The pattern of NOAC usage will be also analyzed descriptively by the following subgroups, if a minimum of 50 patients have been included in the required subgroups:

- Sex (female, male)
- Age at the time of the study visit (75-79, 80-84,  $\geq$ 85 years)
- Comorbidities at the time of the study visit: heart failure, coronary artery disease, peripheral vascular disease, diabetes, chronic kidney disease, liver disease and cancer.

# 14.2 Secondary Outcomes

#### 14.2.1 Patient's characteristics

Patient's characteristics at the time of the study visit by the NOAC type that the patient is taking at the time of the study visit. Patients will be also stratified by the duration since the

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018




first NOAC initiation date until the study visit date (>4 months / ≤4 months) (See Patient's characteristics: refer to Section 11, Table 3.).

### 14.2.2 OAC treatment management

OAC treatment management (since first NOAC initiation until the study visit date), based on the following variables:

- Previous vitamin K antagonist (VKA) treatment (yes/no), VKA treatment duration in years
- Duration since NVAF diagnosis until first NOAC initiation,
- Duration of first NOAC treatment (first NOAC active substance, start and stop date, first NOAC dose and its dose changes),
- Switch to new NOAC (active substance, start/stop date, dose and dose changes, reason for switch to new NOAC): number of patients that switch their first or further NOAC and mean number of switches.
- Total time in NOAC treatment
- History and current antiplatelet treatment (yes/no, start date, end date, active substance).

Patients will be also stratified by the duration since the first NOAC initiation date until the study visit date (> 4 months /  $\leq$ 4 months).

# 14.2.3 Clinical Frailty Scale

Clinical Frailty Scale grading at the time of the study visit, by current NOAC type.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




# 14.2.4 Prevention strategy

The first NOAC usage by NOAC type, for primary prevention or secondary prevention, at the time of first NOAC initiation.

## 14.3 Analysis of Secondary Outcomes

All analysis of secondary outcomes will be performed for the FAS.

#### 14.3.1 Patient's characteristics

Patient's characteristics at the time of the study visit will be summarized descriptively by current NOAC type. Patients will be also stratified by duration since the first NOAC initiation until the study visit date (>4 months / ≤4 months). All covariates related to patient's characteristics (refer to Section 11, Table 3.) will be analyzed descriptively by NOAC type and by the duration since the first NOAC initiation. Standardized differences between Pradaxa® and other NOACs will be estimated for these covariates. For this, a minimum of 50 patients is required for each group.

#### 14.3.2 OAC treatment management

For OAC treatment management, descriptive analysis of previous VKA treatment (yes/no), VKA treatment duration in years, first NOAC treatment duration, first NOAC dose and dose changes, new NOAC treatment duration, new NOAC dose and dose changes. Duration since NVAF diagnosis until first NOAC initiation and total time in NOAC treatment will be described. Also, the reason for switches, the number of patients that switched their first or further NOAC and mean number of switches will be presented. Antiplatelet use will be also summarized.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




The subgroup analysis of these outcomes by the duration since the first NOAC initiation until the study visit date (> 4 months) will also be performed. For this subgroup analysis, a minimum of 50 patients is required for each group.

### 14.3.3 Clinical Frailty Scale

Clinical Frailty Scale grading at the time of the study visit by current NOAC type will be described as the number of patients on each category of frailty as evaluated by the investigator according to patient's records. In addition, CFS score will be summarized in the following two categories: Frailty patients (CFS scoring >4) and Non-frailty patients (CFS scoring ≤4).

## 14.3.4 Prevention strategy

First NOAC usage will be described by NOAC type, for primary prevention or secondary prevention, at the time of first NOAC initiation.



Document:

 $\label{lem:hammanagement-BI} H: \label{lem:hammanagement-BI} H: \label{lem:hammanagement-BI}$ 

AP\_REBELD\_version1.0\_08072020.docx

Author:


Template No.: RWI TP BIOS0013 Revision 1

Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to





Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




#### 14.6 Exploratory analysis

History and current antiplatelet treatment will be described by current NOAC type.

Treatment received at the time of thromboembolic and bleeding events will be described, including NOAC, VKA and antiplatelet treatments.

Doses of current NOAC treatment received by the patient will be described according to HAS-BLED score (as low, intermediate and high risk).

The percentage of underdosed and overdosed patients for current NOAC treatment will be described.

HAS-BLED total score (as  $<3, 3-5, \ge 5$ ) will be described according to NOAC and antiplatelet current treatment.

Multivariate logistic regression will be used to evaluate the association between the Clinical Frailty Scale (dependent variable: Frailty patients - CFS scoring >4 vs Non-frailty patients - CFS scoring ≤4) and the thromboembolic and the bleeding events (independent variables). To calculate this analysis, only events that have occurred subsequent to the start of anticoagulant therapy (not those prior to the start of VKA / NOACs) will be considered. Other factors will be age, sex, BMI, smoking habit, alcohol consumption, time since NVAF diagnosis, NVAF type, modified EHRA scale, procedures and interventions, comorbidity Charlson index and clinical risk factors. Univariate analysis will be performed. All variables which have a P value of less than 0.1 will be included in the multivariate analysis.

#### 15. SAFETY

All outputs for safety analysis will be based on the Safety Analysis Set.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




#### 15.1 Adverse Drug Reactions

The percentage of patients experiencing Adverse Drug Reactions related with BI product Pradaxa®, will be presented. Number and percentage of patients reporting each type of ADRs (SOC and PT) will be reported. ADRs will be described according to type, duration (days), seriousness, reason for seriousness and outcome. Adverse Drug Reaction term (open string variable) will be coded using Medical Dictionary for Regulatory Activities (MedDRA) central coding dictionary, the latest version available.

## 15.2 Serious Adverse Drug Reactions

Serious Adverse Drug Reactions (SADRs) are those ADRs recorded as "Serious" on the Adverse Events page of the (e)CRF. A summary of SADRs by SOC and PT will be prepared.

The percentage of patients experiencing serious related drug reactions (SADRs) with Pradaxa® will be presented. Number and percentage of patients reporting each type of SADRs will be reported.

#### 15.3 Deaths

If any subjects die during Pradaxa® treatment, recorded on the "results in death" or outcome of event" as "fatal" on the (e)CRF, the information will be presented in a summary table and a data listing.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




#### 16. REFERENCES

- Pablo Díez-Villanueva, Albert Arizá -Solé, María Teresa Vidán et al.
   Recommendations of the Geriatric Cardiology Section of the Spanish Society of Cardiology for the Assessment of Frailty in Elderly Patients With Heart Disease.

   Rev Esp Cardiol. 2019;72(1):63–71.
- 3. Camm AJ, Lip GYH, de Caterina R, Savelieva I, Atar D, Hohnloser SH, et al. 2012 focused update of the ESC Guidelines for the management of atrial fibrillation. An update of the 2010 ESC Guidelines for the management of atrial fibrillation developed with the special contribution of the European Heart Rhythm Association Authors/Task Force Members. Eur Heart J. 2012;33:2719-47.
- 4. Kirchhof et al 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. European Heart Journal (2016) 37, 2893–2962.
- 5. Villar R, Meijide H, Castelo L, Mema A, Serrano J, Vares Ma, Ramos V. Escalas en práctica clínica: cardiología. Galicia Clin 2010; 71 (1): 31-36.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




- 6. Charlson M, Szatrowski TP, Peterson J, Gold J (1994) Validation of a combined comorbidity index. J Clin Epidemiol 47: 1245–1251.
- 7. Hosten AO. BUN and Creatinine. In: Walker HK, Hall WD, Hurst JW, editors. Clinical Methods: The History, Physical, and Laboratory Examinations. 3rd ed. Butterworths; Boston: 1990.
- Savino JA 3rd, Halperin JL. Should Patients With Atrial Fibrillation and 1 Stroke Risk Factor (CHA2DS2-VASc Score 1 in Men, 2 in Women) Be Anticoagulated? The CHA2 DS2-VASc 1 Conundrum: Decision Making at the Lower End of the Risk Spectrum. Circulation. 2016 Apr;133(15):1504–11
- 9. Lip G.Y., Banerjee A., Lagrenade I., Lane D.A., Taillandier S., Fauchier L. (2012) Assessing the risk of bleeding in patients with atrial fibrillation: the Loire Valley Atrial Fibrillation Project. Circ Arrhythm Electrophysiol 5:941–948.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




#### 17. APPENDIX 1. MOCK TABLES

## 17.1 Eligibility

Table 5. Eligibility criteria – Patients in the FAS

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total |
|---|---|---|---|---|---|---|
| Total enrolled patients | | | | | | |
| Eligible patients | Eligible patients (FAS) | | | | | |
| | Non-Eligible patients | | | | | |
| Reasons for non-<br>eligible patients | Inclusion criteria 1 | | | | | |
| | Inclusion criteria 2 | | | | | |

Table 6. Main stratification variables

| | | Total |
|---|---|---|
| Total eligible (FAS) | | |
| NOAC type at study visit | Total<br>Dabigatran<br>Rivaroxaban<br>Apixaban<br>Edoxaban | |
| Duration since the first NOAC initiation date until the study visit | <pre>&lt;4 months &gt; 4 months</pre> | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




#### 17.2 Patient's characteristics

Total column will include description of total eligible sample (FAS).

## 17.2.1 Patient's characteristics according to current NOAC type

Table 7. Socio-demographic variables and habits according to current NOAC type

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa® vs<br>others) |
|---|---|---|---|---|---|---|---|
| Age | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Age group | Valid N<br>75-79 years<br>80-84 years<br>≥85 years<br>N missing | | | | | | |
| Sex | Valid N<br>Male, n (%)<br>Female, n (%)<br>N missing | | | | | | |
| Weight (Kg) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Weight (Kg) cat | Valid N<br>≤60 kg, n (%)<br>>60 kg, n (%)<br>N missing | | | | | | |
| Height (cm) | Valid N<br>Mean (SD) | | | | | | |

 $\label{lem:bocument: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S$ 

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa® vs<br>others) |
|---|---|---|---|---|---|---|---|
| | Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| BMI (Kg/m2) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| BMI cat | Valid N Underweight: BMI< 18.5 kg/m2 Normal weight: 18.5 kg/m2<= BMI<= 25 kg/m2 Overweight: 25 kg/m2< BMI<= 30 kg/m2 Obese: 30 kg/m2 <bmi<= 35="" bmi="" kg="" m2="" obese:="" severely=""> 35 kg/m2 N missing</bmi<=> | | | | | | |
| Caregiver | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Place where patients is living | Valid N Home alone At home with partner/other family member/a friend Other's home (e.g. family member's) Nursing home N missing | | | | | | |
| Smoking habit | Valid N<br>Ex-smoker | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

 $AP\_REBELD\_version 1.0\_08072020. docx$ 


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa® vs<br>others) |
|---|---|---|---|---|---|---|---|
| | Smoker<br>Non-smoker<br>N missing | | | | | | |
| Alcohol<br>consumption | Valid N Casual Habitual Abuse Dependence N missing | | | | | | |

Table 8. Analytical laboratory results from the last available blood sample analysis according to current NOAC type

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa® vs<br>others) |
|---|---|---|---|---|---|---|---|
| Serum creatinine (mg/dl) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Serum creatinine<br>Normal levels:<br>0.6-1.2 mg/dl in males<br>0.5-1.1 mg/dl in females | Valid N<br>Normal levels<br>High/low level<br>N missing | | | | | | |
| Creatinine clearance (ml/min) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Creatinine clearance (ml/min): Cockcroft and Gault formula | Valid N<br>Mean (SD)<br>Median (Q1-Q3) | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa® vs<br>others) |
|---|---|---|---|---|---|---|---|
| | Min-Max<br>N missing | | | | | | |
| Creatinine clearance – range (ml/min/1.73m²) | Valid N<br><15<br>15-29<br>30-59<br>60-89<br>≥90<br>N missing | | | | | | |
| AST (UI/L) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| AST<br>Normal values : 7-55 UI/L | Valid N<br>Normal value<br>High/low value<br>N missing | | | | | | |
| ALT (UI/L) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| ALT<br>Normal values: 8-48 UI/L | Valid N<br>Normal value<br>High/low value<br>N missing | | | | | | |
| Total bilirubin (mg/dl) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Total bilirubin<br>Normal values: 0.2-1.2<br>mg/dl | Valid N<br>Normal value<br>High/low value | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

 $AP\_REBELD\_version 1.0\_08072020. docx$ 


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa® vs<br>others) |
|---|---|---|---|---|---|---|---|
| | N missing | | | | | | |
| Haemoglobin (g/dl) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Haemoglobin<br>Normal values: 12-18 g/dl | Valid N<br>Normal value<br>High/low value<br>N missing | | | | | | |
| Platelet levels (x10 <sup>3</sup> /μL) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Platelet<br>Normal values: 150 – 450<br>x103/μL | Valid N<br>Normal value<br>High/low value<br>N missing | | | | | | |

Table 9. NVAF variables according to current NOAC type

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa® vs others) |
|---|---|---|---|---|---|---|---|
| Years since NVAF | Valid N | | | | | | |
| diagnosis | Mean (SD) | | | | | | |
| | Median (Q1-Q3) | | | | | | |
| | Min-Max | | | | | | |
| | N missing | | | | | | |
| Years since NVAF | Valid N | | | | | | |
| diagnosis (patients treated | Mean (SD) | | | | | | |
| previously with VKA) | Median (Q1-Q3) | | | | | | |
| | Min-Max | | | | | | |
| | N missing | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa® vs others) |
|---|---|---|---|---|---|---|---|
| Years since NVAF | Valid N | | | | | | |
| diagnosis (patients treated | Mean (SD) | | | | | | |
| with NOAC as first | Median (Q1-Q3) | | | | | | |
| anticoagulant) | Min-Max | | | | | | |
| | N missing | | | | | | |
| Type of NVAF | Valid N | | | | | | |
| | Persistent | | | | | | |
| | Long standing | | | | | | |
| | persistent | | | | | | |
| | Permanent | | | | | | |
| | Paroxysmal | | | | | | |
| | N missing | | | | | | |
| Modified EHRA scale for | Valid N | | | | | | |
| AF related symptoms | 1-none | | | | | | |
| 1 | 2a-mild | | | | | | |
| | 2b-moderate | | | | | | |
| | 3-severe | | | | | | |
| | 4-disabling | | | | | | |
| | N missing | | | | | | |

Table 10. Procedures and interventions according to current NOAC type

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others) |
|---|---|---|---|---|---|---|---|
| Cardioversion | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Ablation | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Coronary interventions | Valid N<br>No | | | | | | |

Document:

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others) |
|---|---|---|---|---|---|---|---|
| | Yes | | | | | | |
| | N missing | | | | | | |
| Type of coronary | Valid N | | | | | | |
| interventions | Percutaneous coronary intervention | | | | | | |
| | Coronary artery bypass grafting | | | | | | |
| | N missing | | | | | | |
| Pacemaker carrier | Valid N | | | | | | |
| | No | | | | | | |
| | Yes | | | | | | |
| | N missing | | | | | | |

Table 11. Clinical risk factors according to current NOAC type

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| Heart failure | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| NYHA<br>classification | Valid N A - No objective evidence of cardiovascular disease B - Objective evidence of minimal cardiovascular disease C - Objective evidence of moderately severe cardiovascular disease D - Objective evidence of severe cardiovascular disease N missing | | | | | | |
| Left ventricular ejection fraction (%) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| | N missing | | | | | | |
| Coronary<br>artery disease | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Sleep apnoea-<br>hypopnoea<br>syndrome | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Hypertension | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Hyperlipidemia | Valid N<br>No<br>Yes<br>N missing | | | | | | |

Table 12. Charlson Comorbidity Index according to current NOAC type

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| Myocardial infarction | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Congestive heart failure | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Peripheral vascular disease | Valid N<br>No | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| | Yes<br>N missing | | | | | | |
| Cerebrovascular disease | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Dementia | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| COPD | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Connective tissue disease | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Peptic ulcer disease | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Liver disease | Valid N<br>Mild<br>Moderate to<br>severe<br>N missing | | | | | | |
| Diabetes mellitus | Valid N<br>Uncomplicated<br>End-organ<br>damage<br>N missing | | | | | | |
| Hemiplegia | Valid N<br>No<br>Yes | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| | N missing | | | | | | |
| Moderate to severe renal disease | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Solid tumor | Valid N<br>Localized<br>Metastasic<br>N missing | | | | | | |
| Leukemia | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Lymphoma | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| AIDS | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Age-adjusted Charlson<br>Comorbidity index score | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




Table 13. History of thromboembolic events according to current NOAC type

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| History of thromboembolic events | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of total<br>thromboembolic events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| TIA | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of TIA | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Ischemic stroke | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of ischemic strokes | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Hemorrhagic stroke | Valid N<br>No<br>Yes<br>N missing | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| Number of hemorrhagic strokes | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Embolism systemic | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of embolism systemic | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Deep vein thrombosis | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of deep vein thrombosis | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Pulmonary embolism | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of pulmonary embolisms | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Stable angina | Valid N<br>No<br>Yes | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

 $AP\_REBELD\_version 1.0\_08072020. docx$ 


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| | N missing | | | | | | |
| Number of stable anginas | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Unstable angina | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of unstable anginas | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Myocardial infarction with ST segment elevation | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of myocardial infarctions with ST segment elevation | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Myocardial infarction without ST segment elevation | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of myocardial infarctions without ST segment elevation | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




Table 14. History of bleeding events according to current NOAC type

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| History of bleeding events | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of total<br>bleeding events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Intracranial | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of intracranial events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Digestive | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of digestive events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Genitourinary | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of genitourinary events | Valid N<br>Mean (SD) | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| | Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Gingival | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of gingival events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Nasal | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of nasal events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Pulmonary | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number of pulmonary events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Articular-muscular | Valid N<br>No<br>Yes<br>N missing | | | | | | |

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| Number of articular-<br>muscular events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |
| Conjunctival | Valid N<br>No<br>Yes<br>N missing | | | | | | |
| Number conjunctival events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | | |

# Table 15. Risk of stroke (CHA2DS2-VASc) and risk of major bleeding (HAS-BLED) according to current NOAC type

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| CHA2DS2- | Valid N | | | | | | |
| VASc score | Mean (SD) | | | | | | |
| | Median (Q1-Q3)<br>Min-Max | | | | | | |
| | N missing | | | | | | |
| CHA 2DC2 | | | | | | | |
| CHA2DS2- | Valid N | | | | | | |
| VASc (risk | Low risk (score 0 in male; 1 in | | | | | | |
| of stroke) | female) | | | | | | |
| | Moderate risk (score 1 in male; | | | | | | |
| | 2 in female)<br>High risk (score $\geq 2$ in male; $\geq 3$ | | | | | | |
| | in female) $ SCOTe \ge 2$ in male, $ SCOTe \le 2$ | | | | | | |
| | N missing | | | | | | |

Document:

AP\_REBELD\_version1.0\_08072020.docx

Author:


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to

and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| HAS-BLED | Valid N | | | | | | |
| score | Mean (SD) | | | | | | |
| | Median (Q1-Q3) | | | | | | |
| | Min-Max | | | | | | |
| | N missing | | | | | | |
| HAS-BLED | Valid N | | | | | | |
| (risk of | Low risk (score 0) | | | | | | |
| bleeding) | Intermediate risk (score 1-2) | | | | | | |
| | High risk (score ≥3) | | | | | | |
| | N missing | | | | | | |

Table 16. Concomitant treatments to NOAC at study visit according to current NOAC type

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| ARB or ACE inhibitor | No<br>Yes<br>N | | | | | | |
| Beta-blocker | missing Valid N No Yes N | | | | | | |
| Calcium channel<br>blockers | wissing Valid N No Yes N missing | | | | | | |
| Diuretics | Valid N<br>No<br>Yes | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| | N<br>missing | | | | | | |
| Amiodarone | Valid N<br>No<br>Yes<br>N<br>missing | | | | | | |
| Statin | Valid N<br>No<br>Yes<br>N<br>missing | | | | | | |
| Proton pump inhibitor | Valid N<br>No<br>Yes<br>N<br>missing | | | | | | |
| H2-receptor antagonist | | | | | | | |
| Digoxin | Valid N<br>No<br>Yes<br>N<br>missing | | | | | | |
| NSAIDs | Valid N<br>No<br>Yes<br>N<br>missing | | | | | | |
| Dronedarone | Valid N<br>No<br>Yes | | | | | | |

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total | Standardized<br>differences<br>(Pradaxa®<br>vs others |
|---|---|---|---|---|---|---|---|
| | N<br>missing | | | | | | |
| Ketoconazole | Valid N<br>No<br>Yes<br>N<br>missing | | | | | | |
| Cyclosporine | Valid N<br>No<br>Yes<br>N<br>missing | | | | | | |
| Itraconazole | Valid N<br>No<br>Yes<br>N<br>missing | | | | | | |
| Other antiarrhythmics | Valid N<br>No<br>Yes<br>N<br>missing | | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




#### 17.2.2 Patient's characteristics according to duration since the first NOAC initiation

Table 17. Socio-demographic variables and habits according to duration since the first NOAC initiation

| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| Age | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Age group | Valid N 75-79 years 80-84 years ≥85 years N missing | | | |
| Sex | Valid N Male, n (%) Female, n (%) N missing | | | |
| Weight (Kg) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Weight (Kg) cat | Valid N<br>≤60 kg, n (%)<br>>60 kg, n (%)<br>N missing | | | |
| Height (cm) | Valid N Mean (SD) Median (Q1-Q3) Min-Max N missing | | | |
| BMI (Kg/m2) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| BMI cat | Valid N Underweight: BMI< 18.5 kg/m2 Normal weight: 18.5 kg/m2<= BMI<= 25 kg/m2 Overweight: 25 kg/m2< BMI<= 30 kg/m2 Obese: 30 kg/m2 <bmi<= 35="" bmi="" kg="" m2="" obese:="" severely=""> 35 kg/m2 N missing</bmi<=> | | | |
| Caregiver | Valid N<br>No<br>Yes<br>N missing | | | |
| Place where patient is living | Valid N Home alone At home with partner/other family member/a friend Other's home (e.g. family member's) Nursing home N missing | | | |
| Smoking habit | Valid N Ex-smoker Smoker Non-smoker N missing | | | |
| Alcohol<br>consumption | Valid N Casual Habitual Abuse Dependence N missing | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




## Table 18. Analytical laboratory results from the last available blood sample analysis according to duration since the first NOAC initiation

| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| Serum creatinine (mg/dl) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Serum creatinine Normal levels: 0.6-1.2 mg/dl in males 0.5-1.1 mg/dl in females | Valid N<br>Normal levels<br>High/low level<br>N missing | | | |
| Creatinine clearance (ml/min) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Creatinine clearance (ml/min): Cockcroft and Gault formula | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Creatinine clearance – range (ml/min/1.73m <sup>2</sup> ) | Valid N<br><15<br>15-29<br>30-59<br>60-89<br>≥90<br>N missing | | | |
| AST (UI/L) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| AST<br>Normal values: 7-55 UI/L | Valid N<br>Normal value<br>High/low value | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| | N missing | | | |
| ALT (UI/L) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| ALT<br>Normal values: 8-48 UI/L | Valid N<br>Normal value<br>High/low value<br>N missing | | | |
| Total bilirubin (mg/dl) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Total bilirubin<br>Normal values: 0.2-1.2<br>mg/dl | Valid N<br>Normal value<br>High/low value<br>N missing | | | |
| Haemoglobin (g/dl) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Haemoglobin<br>Normal values: 12-18 g/dl | Valid N<br>Normal value<br>High/low value<br>N missing | | | |
| Platelet levels (xμL) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Platelet levels Normal values: $150-450$ $\times 10^3/\mu L$ | Valid N<br>Normal value<br>High/low value<br>N missing | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

 $AP\_REBELD\_version 1.0\_08072020. docx$ 


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




Table 19. NVAF variables according to duration since the first NOAC initiation

| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| Years since NVAF diagnosis | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Years since NVAF diagnosis (patients treated previously with VKA) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Years since NVAF diagnosis<br>(patients treated with NOAC<br>as first anticoagulant) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Type of NVAF | Valid N Persistent Long standing persistent Permanent Paroxysmal N missing | | | |
| Modified EHRA scale for AF related symptoms | Valid N 1-none 2a-mild 2b-moderate 3-severe 4-disabling N missing | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




Table 20. Procedures and interventions according to duration since the first NOAC initiation

| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| Cardioversion | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| Ablation | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| Coronary interventions | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| Type of coronary | Valid N | | | |
| interventions | Percutaneous coronary | | | |
| | intervention | | | |
| | Coronary artery bypass grafting | | | |
| | N missing | | | |
| Pacemaker carrier | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |

Table 21. Clinical risk factors according to duration since the first NOAC initiation

| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| Heart failure | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| NYHA | Valid N | | | |
| classification | A - No objective evidence of cardiovascular | | | |
| | disease | | | |
| | B - Objective evidence of minimal | | | |
| | cardiovascular disease | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| | C - Objective evidence of moderately severe cardiovascular disease D - Objective evidence of severe cardiovascular disease | | | · |
| | N missing | | | |
| Left ventricular ejection fraction (%) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Coronary<br>artery disease | Valid N<br>No<br>Yes<br>N missing | | | |
| Sleep apnoea-<br>hypopnoea<br>syndrome | Valid N<br>No<br>Yes<br>N missing | | | · |
| Hypertension | Valid N<br>No<br>Yes<br>N missing | | | |
| Hyperlipidemia | Valid N<br>No<br>Yes<br>N missing | | | |

Table 22. Comorbidity Charlson Index according to duration since the first NOAC initiation

| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| Myocardial infarction | Valid N<br>No<br>Yes<br>N missing | | | |
| Congestive heart failure | Valid N<br>No<br>Yes | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to

<sup>.</sup> and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| | N missing | | | |
| Peripheral vascular disease | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| Cerebrovascular disease | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| Dementia | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| COPD | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| Connective tissue disease | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| Peptic ulcer disease | Valid N | | | |
| - | No | | | |
| | Yes | | | |
| | N missing | | | |
| Liver disease | Valid N | | | |
| | Mild | | | |
| | Moderate to | | | |
| | severe | | | |
| | N missing | | | |
| Diabetes mellitus | Valid N | | | |
| | Uncomplicated | | | |
| | End-organ damage | | | |
| | N missing | | | |
| Hemiplegia | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| Moderate to severe renal disease | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| Solid tumor | Valid N | | | |
| | Localized | | | |
| | Metastasic | | | |
| | N missing | | | |
| Leukemia | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| Lymphoma | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| AIDS | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| Age-adjusted Charlson | Valid N | | | |
| Comorbidity index score | Mean (SD) | | | |
| | Median (Q1-Q3) | | | |
| | Min-Max | | | |
| | N missing | | | |

Table 23. History of thromboembolic events according to duration since the first NOAC initiation

| | | ≤4 months | >4 months | Total |
|-----------------------|----------------|-----------|-----------|-------|
| History of | Valid N | | | |
| thromboembolic events | No | | | |
| | Yes | | | |
| | N missing | | | |
| Number of total | Valid N | | | |
| thromboembolic events | Mean (SD) | | | |
| | Median (Q1-Q3) | | | |
| | Min-Max | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| | N missing | | | |
| TIA | Valid N<br>No<br>Yes<br>N missing | | | |
| Number of TIA | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Ischemic stroke | Valid N<br>No<br>Yes<br>N missing | | | |
| Number of ischemic strokes | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Hemorrhagic stroke | Valid N<br>No<br>Yes<br>N missing | | | |
| Number of hemorrhagic strokes | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Embolism systemic | Valid N<br>No<br>Yes<br>N missing | | | |
| Number of embolism systemic | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Deep vein thrombosis | Valid N | | | |

Document:

 $\label{lem:hamman} \mbox{H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\SAP\SAP\BOOTO\BO$ 

AP\_REBELD\_version1.0\_08072020.docx

Author:


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| | No<br>Yes<br>N missing | | | |
| Number of deep vein thrombosis | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Pulmonary embolism | Valid N<br>No<br>Yes<br>N missing | | | |
| Number of pulmonary embolisms | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Stable angina | Valid N<br>No<br>Yes<br>N missing | | | |
| Number of stable anginas | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Unstable angina | Valid N<br>No<br>Yes<br>N missing | | | |
| Number of unstable anginas | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Myocardial infarction with ST segment elevation | Valid N<br>No<br>Yes | | | |

Document:

H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx

Author:


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to



| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| | N missing | | | |
| Number of myocardial infarctions with ST segment elevation | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Myocardial infarction without ST segment elevation | Valid N<br>No<br>Yes<br>N missing | | | |
| Number of myocardial infarctions without ST segment elevation | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

Table 24. History of bleeding events according to duration since the first NOAC initiation

| | | ≤4 months | >4 months | Total |
|--------------------------|----------------|-----------|-----------|-------|
| History of bleeding | Valid N | | | |
| events | No | | | |
| | Yes | | | |
| | N missing | | | |
| Number of total bleeding | Valid N | | | |
| events | Mean (SD) | | | |
| | Median (Q1-Q3) | | | |
| | Min-Max | | | |
| | N missing | | | |
| Intracranial | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| Number of intracranial | Valid N | | | |
| events | Mean (SD) | | | |
| | Median (Q1-Q3) | | | |
| | Min-Max | | | |
| | N missing | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to

<sup>.</sup> and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| Digestive | Valid N<br>No<br>Yes<br>N missing | | | |
| Number of digestive events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Genitourinary | Valid N<br>No<br>Yes<br>N missing | | | |
| Number of genitourinary events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Gingival | Valid N<br>No<br>Yes<br>N missing | | | |
| Number of gingival events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Nasal | Valid N<br>No<br>Yes<br>N missing | | | |
| Number of nasal events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Pulmonary | Valid N<br>No | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| | Yes<br>N missing | | | |
| Number of pulmonary events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Articular-muscular | Valid N<br>No<br>Yes<br>N missing | | | |
| Number of articular-<br>muscular events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Conjunctival | Valid N<br>No<br>Yes<br>N missing | | | |
| Number conjunctival events | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

# Table 25. Risk of stroke (CHA2DS2-VASc) and risk of major bleeding (HAS-BLED) according to duration since the first NOAC initiation

| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| CHA2DS2-VASc score | Valid N | | | |
| | Mean (SD) | | | |
| | Median (Q1-Q3) | | | |
| | Min-Max | | | |
| | N missing | | | |
| CHA2DS2-VASc (risk of | Valid N | | | |
| stroke) | Low risk (score 0 in male; 1 in female) | | | |

Document:

 $\label{thm:hamman} \mbox{H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\SAP\SAP\BOX - BI\Proyecto\Estadistica\SAP\SAP\SAP\BOX - BI\Proyecto\BOX - BI\Proyecto\BO$ 

AP\_REBELD\_version1.0\_08072020.docx

Author:


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| | Moderate risk (score 1 in male; 2 in female) High risk (score ≥2 in male; ≥3 in female) N missing | | | |
| HAS-BLED score | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| HAS-BLED (risk of bleeding) | Valid N Low risk (score 0) Intermediate risk (score 1-2) High risk (score ≥3) N missing | | | |

Table 26. Concomitant treatments to NOAC at study visit according to duration since the first NOAC initiation

| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| ARB or ACE inhibitor | Valid N<br>No<br>Yes<br>N missing | | | |
| Beta-blocker | Valid N<br>No<br>Yes<br>N missing | | | |
| Calcium<br>channel<br>blockers | Valid N<br>No<br>Yes<br>N missing | | | |
| Diuretics | Valid N<br>No<br>Yes<br>N missing | | | |
| Amiodarone | Valid N<br>No | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| | Yes<br>N missing | | | |
| Statin | Valid N<br>No<br>Yes<br>N missing | | | |
| Proton pump inhibitor | Valid N<br>No<br>Yes<br>N missing | | | |
| H2-receptor antagonist | Valid N<br>No<br>Yes<br>N missing | | | |
| Digoxin | Valid N<br>No<br>Yes<br>N missing | | | |
| NSAIDs | Valid N<br>No<br>Yes<br>N missing | | | |
| Dronedarone | Valid N<br>No<br>Yes<br>N missing | | | |
| Ketoconazole | Valid N<br>No<br>Yes<br>N missing | | | |
| Cyclosporine | Valid N<br>No<br>Yes<br>N missing | | | |
| Itraconazole | Valid N<br>No<br>Yes<br>N missing | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | ≤4 months | >4 months | Total |
|-----------------|-----------|-----------|-----------|-------|
| | Valid N | | | |
| antiarrhythmics | No<br>Yes | | | |
| | N missing | | | |

# 17.3 Outcomes

# 17.3.1 Primary outcome: Current NOAC

Table 27. Type of NOAC, dose and duration since first NOAC initiation at study visit according to sex

| | | Male | Female | Total |
|---|---|---|---|---|
| Current NOAC | Valid N<br>Dabigatran<br>Rivaroxaban<br>Apixaban | | | |
| | Edoxaban<br>N missing | | | |
| Dabigatran dose | Valid N<br>110mg BID<br>150mg BID<br>N missing | | | |
| Rivaroxaban dose | Valid N<br>15mg QD<br>20mg QD<br>N missing | | | |
| Apixaban dose | Valid N<br>2.5mg BID<br>5mg BID<br>N missing | | | |
| Edoxaban dose | Valid N<br>30mg QD<br>60mg QD<br>N missing | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Male | Female | Total |
|---|---|---|---|---|
| Years since first NOAC initiation to study visit | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

BDI: twice a day; QD: once a day

Table 28. Type of NOAC, dose and duration since fist NOAC initiation at study visit according to age

| | | 75-79<br>years | 80-84<br>years | ≥85 years | Total |
|---|---|---|---|---|---|
| Current NOAC | Valid N Dabigatran Rivaroxaban Apixaban Edoxaban N missing | | | | |
| Dabigatran dose | Valid N<br>110mg BID<br>150mg BID<br>N missing | | | | |
| Rivaroxaban dose | Valid N<br>15mg QD<br>20mg QD<br>N missing | | | | |
| Apixaban dose | Valid N<br>2.5mg BID<br>5mg BID<br>N missing | | | | |
| Edoxaban dose | Valid N<br>30mg QD<br>60mg QD<br>N missing | | | | |
| Years since first NOAC initiation to study visit | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | 75-79<br>years | 80-84<br>years | ≥85 years | Total |
|-----------|----------------|----------------|-----------|-------|
| N missing | | | | |

BDI: twice a day; QD: once a day

Table 29. Type of NOAC, dose and duration since fist NOAC initiation at study visit according to heart failure

| | | I | Heart failure | |
|---|---|---|---|---|
| | | No | Yes | Total |
| Current NOAC | Valid N Dabigatran Rivaroxaban Apixaban Edoxaban N missing | | | |
| Dabigatran dose | Valid N<br>110mg BID<br>150mg BID<br>N missing | | | |
| Rivaroxaban dose | Valid N<br>15mg QD<br>20mg QD<br>N missing | | | |
| Apixaban dose | Valid N<br>2.5mg BID<br>5mg BID<br>N missing | | | |
| Edoxaban dose | Valid N<br>30mg QD<br>60mg QD<br>N missing | | | |
| Years since first NOAC initiation to study visit | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

BDI: twice a day; QD: once a day

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to

and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




Table 30. Type of NOAC, dose and duration since fist NOAC initiation at study visit according to coronary artery disease

| | | Coronary artery disease | | |
|---|---|---|---|---|
| | | No | Yes | Total |
| Current NOAC | Valid N Dabigatran Rivaroxaban Apixaban Edoxaban N missing | | | |
| Dabigatran dose | Valid N<br>110mg BID<br>150mg BID<br>N missing | | | |
| Rivaroxaban dose | Valid N<br>15mg QD<br>20mg QD<br>N missing | | | |
| Apixaban dose | Valid N<br>2.5mg BID<br>5mg BID<br>N missing | | | |
| Edoxaban dose | Valid N<br>30mg QD<br>60mg QD<br>N missing | | | |
| Years since first NOAC initiation to study visit | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

BDI: twice a day; QD: once a day

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




Table 31. Type of NOAC, dose and duration since fist NOAC initiation at study visit according to peripheral vascular disease

| | | Peripher | ral vascular d | lisease |
|---|---|---|---|---|
| | | No | Yes | Total |
| Current NOAC | Valid N Dabigatran Rivaroxaban Apixaban Edoxaban N missing | | | |
| Dabigatran dose | Valid N<br>110mg BID<br>150mg BID<br>N missing | | | |
| Rivaroxaban dose | Valid N<br>15mg QD<br>20mg QD<br>N missing | | | |
| Apixaban dose | Valid N<br>2.5mg BID<br>5mg BID<br>N missing | | | |
| Edoxaban dose | Valid N<br>30mg QD<br>60mg QD<br>N missing | | | |
| Years since first NOAC initiation to study visit | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

BDI: twice a day; QD: once a day

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




Table 32. Type of NOAC, dose and duration since fist NOAC initiation at study visit according to diabetes

| | | | Diabetes | |
|---|---|---|---|---|
| | | No | Yes | Total |
| Current NOAC | Valid N Dabigatran Rivaroxaban Apixaban Edoxaban N missing | | | |
| Dabigatran dose | Valid N<br>110mg BID<br>150mg BID<br>N missing | | | |
| Rivaroxaban dose | Valid N<br>15mg QD<br>20mg QD<br>N missing | | | |
| Apixaban dose | Valid N<br>2.5mg BID<br>5mg BID<br>N missing | | | |
| Edoxaban dose | Valid N<br>30mg QD<br>60mg QD<br>N missing | | | |
| Years since first NOAC initiation to study visit | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

BDI: twice a day; QD: once a day

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




Table 33. Type of NOAC, dose and duration since fist NOAC initiation at study visit according to chronic kidney disease

| | | Chron | ic kidney dis | ease |
|---|---|---|---|---|
| | | No | Yes | Total |
| Current NOAC | Valid N Dabigatran Rivaroxaban Apixaban Edoxaban N missing | | | |
| Dabigatran dose | Valid N<br>110mg BID<br>150mg BID<br>N missing | | | |
| Rivaroxaban dose | Valid N<br>15mg QD<br>20mg QD<br>N missing | | | |
| Apixaban dose | Valid N<br>2.5mg BID<br>5mg BID<br>N missing | | | |
| Edoxaban dose | Valid N<br>30mg QD<br>60mg QD<br>N missing | | | |
| Years since first NOAC initiation to study visit | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

BDI: twice a day; QD: once a day

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




Table 34. Type of NOAC, dose and duration since fist NOAC initiation at study visit according to liver disease

| | | Liver disease | | |
|---|---|---|---|---|
| | | No | Yes | Total |
| Current NOAC | Valid N Dabigatran Rivaroxaban Apixaban Edoxaban N missing | | | |
| Dabigatran dose | Valid N<br>110mg BID<br>150mg BID<br>N missing | | | |
| Rivaroxaban dose | Valid N<br>15mg QD<br>20mg QD<br>N missing | | | |
| Apixaban dose | Valid N<br>2.5mg BID<br>5mg BID<br>N missing | | | |
| Edoxaban dose | Valid N<br>30mg QD<br>60mg QD<br>N missing | | | |
| Years since first NOAC initiation to study visit | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

BDI: twice a day; QD: once a day

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




Table 35. Type of NOAC, dose and duration since fist NOAC initiation at study visit according to cancer

| | | | Cancer | |
|---|---|---|---|---|
| | | No | Yes | Total |
| Current NOAC | Valid N<br>Dabigatran<br>Rivaroxaban<br>Apixaban<br>Edoxaban<br>N missing | | | |
| Dabigatran dose | Valid N<br>110mg BID<br>150mg BID<br>N missing | | | |
| Rivaroxaban dose | Valid N<br>15mg QD<br>20mg QD<br>N missing | | | |
| Apixaban dose | Valid N<br>2.5mg BID<br>5mg BID<br>N missing | | | |
| Edoxaban dose | Valid N<br>30mg QD<br>60mg QD<br>N missing | | | |
| Years since first NOAC initiation to study visit | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |

BDI: twice a day; QD: once a day

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




# 17.3.2 Secondary outcome: OAC treatment management

Table 36. Previous VKA treatment and duration according to duration since the first NOAC initiation

| | | ≤4 months | >4 months | Total |
|---------------------|----------------|-----------|-----------|-------|
| Previous VKA | Valid N | | | |
| | No | | | |
| | Yes | | | |
| | N missing | | | |
| Type of VKA | Valid N | | | |
| | Acenocoumarol | | | |
| | Warfarin | | | |
| | N missing | | | |
| Years with | Valid N | | | |
| Acenocoumarol | Mean (SD) | | | |
| | Median (Q1-Q3) | | | |
| | Min-Max | | | |
| | N missing | | | |
| Years with Warfarin | Valid N | | | |
| | Mean (SD) | | | |
| | Median (Q1-Q3) | | | |
| | Min-Max | | | |
| | N missing | | | |
| Total VKA treatment | Valid N | | | |
| duration in years | Mean (SD) | | | |
| | Median (Q1-Q3) | | | |
| | Min-Max | | | |
| | N missing | | | |

Table 37. Durations since NVAF diagnosis until first NOAC initiation, first NOAC received, first NOAC dose, dose changes and first NOAC treatment duration according to duration since the first NOAC initiation

| | | ≤4 | >4 | Tota | l |
|---|---|---|---|---|---|
| | | months | months | 1 | |
| Months since NVAF diagnosis until first NOAC | Valid N | | | | |
| initiation | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |

Document:

 $\label{lem:hamman} \mbox{H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\SAP\SAP\BOOTO\BO$ 

AP\_REBELD\_version1.0\_08072020.docx

Author:


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | ≤4 months | >4<br>months | Tota<br>1 |
|---|---|---|---|---|
| | Min-Max<br>N missing | | | |
| First NOAC received | Valid N Dabigatran Rivaroxaban Apixaban Edoxaban N missing | | | |
| First NOAC dose: Dabigatran | Valid N<br>110mg BID<br>150mg BID<br>N missing | | | |
| First NOAC dose: Rivaroxaban | Valid N<br>15mg QD<br>20mg QD<br>N missing | | | |
| First NOAC dose: Apixaban | Valid N<br>2.5mg BID<br>5mg BID<br>N missing | | | |
| First NOAC dose: Edoxaban | Valid N<br>30mg QD<br>60mg QD<br>N missing | | | |
| Changes in first NOAC dose | Valid N No Yes (increase) Yes (decrease) N missing | | | |
| First NOAC treatment duration in years* | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Reason for first NOAC treatment discontinuation* | Valid N<br>Lack of effectiveness<br>Investigator decision | | | |

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | ≤4<br>months | >4<br>months | Tota<br>1 |
|---|---|---|---|---|
| | Patient decision<br>Adverse event<br>N missing | | | |
| Reason for first NOAC treatment change dose* | Valid N Lack of effectiveness Investigator decision Patient decision Adverse event N missing | | | |

BDI: twice a day; QD: once a day

Table 38. Number of switches to a new NOAC and reason for switches according to duration since the first NOAC initiation

| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| Number of switches to a | Valid N | | | |
| new NOAC | Mean (SD) | | | |
| | Median (Q1-Q3) | | | |
| | Min-Max | | | |
| | N missing | | | |
| Number of switches to a | Valid N | | | |
| new NOAC | 0 | | | |
| | 1 | | | |
| | 2 | | | |
| | 3 | | | |
| | N missing | | | |
| Switchers | Valid N* | | | |
| | Dabigatran to Rivaroxaban | | | |
| | Dabigatran to Apixaban | | | |
| | Dabigatran to Edoxaban | | | |
| | Rivaroxaban to Dabigatran | | | |
| | Rivaroxaban to Apixaban | | | |
| | Rivaroxaban to Edoxaban | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to

<sup>\*</sup>Only patients who stopped first NOAC treatment

<sup>.</sup> and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| | Apixaban to Dabigatran Apixaban to Rivaroxaban Apixaban to Edoxaban Edoxaban to Dabigatran Edoxaban to Rivaroxaban Edoxaban to Apixaban N missing | | | |
| Reason for switch | Valid N* Lack of effectiveness Investigator's decision Patient's decision Adverse effect N missing | | | |

<sup>\*</sup>Valid N corresponds to the total of switches

Table 39. New NOAC received, new NOAC dose and new NOAC treatment duration according to duration since the first NOAC initiation (SECOND NOAC)

| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| Second NOAC received | Valid N<br>Dabigatran<br>Rivaroxaban<br>Apixaban<br>Edoxaban<br>N missing | | | |
| Second NOAC dose:<br>Dabigatran | Valid N<br>110mg BID<br>150mg BID<br>N missing | | | |
| Second NOAC dose:<br>Rivaroxaban | Valid N<br>15mg QD<br>20mg QD<br>N missing | | | |
| Second NOAC dose:<br>Apixaban | Valid N<br>2.5mg BID<br>5mg BID<br>N missing | | | |

Document:

 $\label{thm:hamman} \mbox{H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\SAP\SAP\BOOTO\BO$ 

AP\_REBELD\_version1.0\_08072020.docx

Author:


Template No.: RWI\_TP\_BIOS0013 Revision 1

Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to

and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




| | | ≤4 months | >4 months | Total |
|---|---|---|---|---|
| Second NOAC dose:<br>Edoxaban | Valid N<br>30mg QD<br>60mg QD<br>N missing | | | |
| Changes in second<br>NOAC dose | Valid N<br>No<br>Yes (increase)<br>Yes (decrease)<br>N missing | | | |
| Second NOAC treatment duration in years* | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | |
| Reason for second<br>NOAC treatment<br>discontinuation* | Valid N Lack of effectiveness Investigator decision Patient decision Adverse event N missing | | | |
| Reason for second<br>NOAC treatment change<br>dose* | Valid N Lack of effectiveness Investigator decision Patient decision Adverse event N missing | | | |

BDI: twice a day; QD: once a day

Table 39. will be repeated for each treatment switch during follow-up.

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to

<sup>\*</sup>Only patients who stopped second NOAC treatment




Table 40. Total time (in years) in NOAC treatment

| | | ≤4 months | >4 months | Total |
|----------------------|-------------|-----------|-----------|-------|
| Total time in NOAC | Valid N | | | |
| treatment (in years) | Mean (SD) | | | |
| | Median (Q1- | | | |
| | Q3) | | | |
| | Min-Max | | | |
| | N missing | | | |
| Total time in NOAC | Valid N | | | |
| treatment (cat) | <1 year | | | |
| | 1-2 years | | | |
| | 2-3 years | | | |
| | >3 years | | | |
| | N missing | | | |

Table 41. History and current antiplatelet treatment according to duration since the first NOAC initiation

| | | ≤4 months | >4 months | Total |
|----------------------------|----------------|-----------|-----------|-------|
| Antiplatelet treatments | Valid N | | | |
| received (all) | Aspirin | | | |
| | Clopidogrel | | | |
| | Prasugrel | | | |
| | Ticlopidine | | | |
| | Ticagrelor | | | |
| | Cilostazol | | | |
| | Triflusal | | | |
| | Dipyridamole | | | |
| | Others | | | |
| | N missing | | | |
| Time in treatment with | Valid N | | | |
| antiplatelet agents (in | Mean (SD) | | | |
| years) | Median (Q1-Q3) | | | |
| | Min-Max | | | |
| | N missing | | | |
| Current antiplatelet | Valid N | | | |
| treatment (at study visit) | None | | | |

Document:

 $\label{thm:hamman} \mbox{H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\SAP\SAP\BOX - BI\Proyecto\Estadistica\SAP\SAP\SAP\BOX - BI\Proyecto\BOX - BI\Proyecto\BO$ 

AP\_REBELD\_version1.0\_08072020.docx

Author:


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | ≤4 months | >4 months | Total |
|--------------|-----------|-----------|-------|
| Aspirin | | | |
| Clopidogrel | | | |
| Prasugrel | | | |
| Ticlopidine | | | |
| Ticagrelor | | | |
| Cilostazol | | | |
| Triflusal | | | |
| Dipyridamole | | | |
| Others | | | |
| N missing | | | |

# 17.3.3 Secondary outcome: Clinical Frailty Scale

Table 42. Clinical Frailty Scale grading at the time of the study visit according to current NOAC type

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total |
|---|---|---|---|---|---|---|
| CFS score | Valid N | | | | | |
| | 1-Very fit | | | | | |
| | 2-Well | | | | | |
| | 3-Managing well | | | | | |
| | 4-Vulnerable | | | | | |
| | 5-Mildly frail | | | | | |
| | 6-Moderately frail | | | | | |
| | 7-Severely frail | | | | | |
| | 8-Very severely frail | | | | | |
| | 9-Terminally ill | | | | | |
| | N missing | | | | | |
| CFS | Valid N | | | | | |
| (categorized) | Non-frailty patients (CFS scoring ≤4) | | | | | |
| | Frailty patients (CFS scoring >4) | | | | | |
| | N missing | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




# 17.3.4 Secondary outcome: Prevention strategy

Table 43. First NOAC usage at the time of first NOAC initiation according to current NOAC type

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total |
|---|---|---|---|---|---|---|
| Reason for prescription of | Valid N | | | | | |
| the first NOAC | Primary prevention | | | | | |
| | Secondary | | | | | |
| | prevention | | | | | |
| | N missing | | | | | |



Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to






# 17.4 Additional tables

Table 45. Historic and current antiplatelet treatment according to current NOAC type

| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total |
|---|---|---|---|---|---|---|
| Antiplatelet treatments | Valid N | | | | | |
| received (all) | Aspirin | | | | | |
| | Clopidogrel | | | | | |
| | Prasugrel | | | | | |
| | Ticlopidine | | | | | |
| | Ticagrelor | | | | | |
| | Cilostazol | | | | | |
| | Triflusal | | | | | |
| | Dipyridamole | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | Total |
|---|---|---|---|---|---|---|
| | Others<br>N missing | | | | | |
| Time in treatment with antiplatelet agents (in years) | Valid N<br>Mean (SD)<br>Median (Q1-Q3)<br>Min-Max<br>N missing | | | | | |
| Current antiplatelet treatment (at study visit) | Valid N None Aspirin Clopidogrel Prasugrel Ticlopidine Ticagrelor Cilostazol Triflusal Dipyridamole Others N missing | | | | | |

Table 46. Treatment received at the moment of thromboembolic events (1st part)

| | | TIA | Ischemic<br>stroke | Hemorrhagic stroke | Embolism<br>systemic | Deep vein thrombosis |
|---|---|---|---|---|---|---|
| Treatment (VKA/NOAC/ antiplatelet) | Valid N* No Yes N missing | | | | | |
| VKA | Valid N* No Yes N missing | | | | | |
| Type of VKA | Valid N<br>Acenocoumarol<br>Warfarin<br>N missing | | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | TIA | Ischemic stroke | Hemorrhagic stroke | Embolism systemic | Deep vein thrombosis |
|---|---|---|---|---|---|---|
| NOAC | Valid N*<br>No<br>Yes<br>N missing | | | | | |
| Type of<br>NOAC | Valid N Dabigatran Rivaroxaban Apixaban Edoxaban N missing | | | | | |
| Antiplatelet | Valid N* No Yes N missing | | | | | |
| Type of antiplatelet | Valid N Aspirin Clopidogrel Prasugrel Ticlopidine Ticagrelor Cilostazol Triflusal Dipyridamole Others N missing | | | | | |

<sup>\*</sup>Number of events in each column.

One event could be associated with more than one treatment

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




Table 47. Treatment received at the moment of thromboembolic events (2<sup>nd</sup> part)

| | | Pulmonary<br>embolism | Stable angina | Unstable<br>angina | Myocardial<br>infarction with<br>ST segment<br>elevation | Myocardial infarction without ST segment elevation |
|---|---|---|---|---|---|---|
| Treatment (VKA/NOAC/ antiplatelet) | Valid N* No Yes N missing | | | | | |
| VKA | Valid N* No Yes N missing | | | | | |
| Type of VKA | Valid N<br>Acenocoumarol<br>Warfarin<br>N missing | | | | | |
| NOAC | Valid N* No Yes N missing | | | | | |
| Type of<br>NOAC | Valid N<br>Dabigatran<br>Rivaroxaban<br>Apixaban<br>Edoxaban<br>N missing | | | | | |
| Antiplatelet | Valid N* No Yes N missing | | | | | |
| Type of antiplatelet | Valid N Aspirin Clopidogrel Prasugrel Ticlopidine Ticagrelor Cilostazol | | | | | |

Document:

H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx

Author:


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | Pulmonary<br>embolism | Stable angina | Unstable<br>angina | Myocardial<br>infarction with<br>ST segment<br>elevation | Myocardial<br>infarction<br>without ST<br>segment<br>elevation |
|---|---|---|---|---|---|
| Triflusal<br>Dipyridamole<br>Others<br>N missing | , | | | | |

<sup>\*</sup>Number of events in each column

One event could be associated with more than one treatment

Table 48. Treatment received at the moment of bleeding events (1st part)

| | | Intracranial | Digestive | Genitourinary | Gingival |
|---|---|---|---|---|---|
| Treatment (VKA/NOAC/ antiplatelet) | Valid N* No Yes N missing | | | | |
| VKA | Valid N* No Yes N missing | | | | |
| Type of VKA | Valid N<br>Acenocoumarol<br>Warfarin<br>N missing | | | | |
| NOAC | Valid N* No Yes N missing | | | | |
| Type of<br>NOAC | Valid N<br>Dabigatran<br>Rivaroxaban<br>Apixaban<br>Edoxaban<br>N missing | | | | |
| Antiplatelet | Valid N* | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Intracranial | Digestive | Genitourinary | Gingival |
|---|---|---|---|---|---|
| | No<br>Yes<br>N missing | | | | |
| Type of antiplatelet | Valid N Aspirin Clopidogrel Prasugrel Ticlopidine Ticagrelor Cilostazol Triflusal Dipyridamole Others N missing | | | | |

<sup>\*</sup>Number of events in each column

One event could be associated with more than one treatment

Table 49. Treatment received at the moment of thromboembolic events (2<sup>nd</sup> part)

| | | Nasal | Pulmonary | Articular-<br>muscular | Conjunctival |
|---|---|---|---|---|---|
| Treatment | Valid N* | | | | |
| (VKA/NOAC/ | No | | | | |
| antiplatelet) | Yes | | | | |
| | N missing | | | | |
| VKA | Valid N* | | | | |
| | No | | | | |
| | Yes | | | | |
| | N missing | | | | |
| Type of VKA | Valid N | | | | |
| | Acenocoumarol | | | | |
| | Warfarin | | | | |
| | N missing | | | | |
| NOAC | Valid N* | · | | | |
| | No | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Nasal | Pulmonary | Articular-<br>muscular | Conjunctival |
|---|---|---|---|---|---|
| | Yes<br>N missing | | | | |
| Type of<br>NOAC | Valid N Dabigatran Rivaroxaban Apixaban Edoxaban N missing | | | | |
| Antiplatelet | Valid N* No Yes N missing | | | | |
| Type of antiplatelet | Valid N Aspirin Clopidogrel Prasugrel Ticlopidine Ticagrelor Cilostazol Triflusal Dipyridamole Others N missing | | | | |

<sup>\*</sup>Number of events in each column

One event could be associated with more than one treatment

Table 50. Current NOAC dose according to HAS-BLED

| | | | HAS-BLED | | |
|---|---|---|---|---|---|
| | | Low risk | Intermediate risk | High<br>risk | Total |
| Dabigatran dose | Valid N<br>110mg BID<br>150mg BID<br>N missing | | | | |
| Rivaroxaban dose | Valid N | | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | | HAS-BLED | | |
|---|---|---|---|---|---|
| | | Low risk | Intermediate risk | High<br>risk | Total |
| | 15mg QD<br>20mg QD<br>N missing | | | | |
| Apixaban dose | Valid N<br>2.5mg BID<br>5mg BID<br>N missing | | | | |
| Edoxaban dose | Valid N<br>30mg QD<br>60mg QD<br>N missing | | | | |

Table 51. Overdosing and underdosing of current NOACs

| | | Appropriately dosed (n,%) | Underdosed (n,%) | Overdosed (n,%) |
|---|---|---|---|---|
| Dabigatran | Dabigatran (Age <80 years) | | | NA |
| | Dabigatran (Age ≥80 years) | | NA | |
| | Dabigatran (75-79 years and HAS-BLED < 3) | | | NA |
| | Dabigatran (75-79 years and HAS-BLED ≥ 3) | | NA | |
| | Dabigatran (creatinine clearance >50mL/min) | | | NA |
| | Dabigatran (creatinine clearance 30-50mL/min) | | NA | |
| Rivaroxaban | Rivaroxaban (creatinine clearance >50mL/min) | | | NA |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | | Appropriately dosed (n,%) | Underdosed (n,%) | Overdosed (n,%) |
|---|---|---|---|---|
| | Rivaroxaban (creatinine clearance ≤50mL/min) | | NA | |
| Apixaban | Apixaban (Age <80 years) | | | NA |
| | Apixaban (Age ≥80 years) | | NA | |
| | Apixaban (Body weight > 60 kg) | | | NA |
| | Apixaban (Body weight ≤ 60 kg) | | NA | |
| | Apixaban (Serum creatinine < 1,5 mg/dl or creatinine clearance ≥30mL/min) | | | NA |
| | Apixaban (Serum creatinine ≥ 1,5 mg/dl or creatinine clearance <30mL/min) | | NA | |
| Edoxaban | Edoxaban (Body weight > 60 kg) | | | NA |
| | Edoxaban (Body weight ≤ 60 kg) | | NA | |
| | Edoxaban (creatinine clearance >50mL/min) | | | NA |
| | Edoxaban (creatinine clearance 15-50mL/min) | | NA | |

Table 52. HAS-BLED score according NOAC+antiplatelet current treatment

| | | | HAS-BLED score | | | |
|---|---|---|---|---|---|---|
| | | Valid N | <3 | 3-5 | ≥5 | N missing |
| Current treatment | Dabigatran+aspirin | | | | | |
| | Dabigatran+clopidogrel | | | | | |
| | Dabigatran+peasugrel | | | | | |
| | (for all combinations) | | | | | |

Row percentage will be calculated

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




Table 53. Multivariate logistic model to evaluate the association between the Clinical Frailty Scale and the thromboembolic and the bleeding events

| Variable | Estimate | Standard<br>error | t-value | Pr> t | OR |
|----------|----------|-------------------|---------|-------|----|

<sup>\*</sup>dependent variable: CFS in two categories: Frailty patients - CFS scoring >4 vs Non-frailty patients - CFS scoring ≤4)

# 17.5 Adverse Drug Reactions

Table 54. Patients with ADRs associated to BI product Pradaxa®

| | | Pradaxa<br>150mg |
|---|---|---|
| ADRs associated to BI product (Pradaxa®) | Total patients<br>No<br>Yes | |
| Type of ADR (multi-response) | SOC1<br>PT11<br>PT12<br><br>SOC2<br>PT21<br>PT22<br> | |
| ADR outcome (multi-response) | Recovered Not yet recovered | |

Document:

AP\_REBELD\_version1.0\_08072020.docx

Author:


Template No.: RWI TP BIOS0013 Revision 1

Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to

<sup>\*</sup>independent variables: thromboembolic and bleeding events. Other factors will be age, sex, BMI, smoking habit, alcohol consumption, time since NVAF diagnosis, NVAF type, modified EHRA scale, procedures and interventions, comorbidity Charlson index and clinical risk factors. Univariate analysis will be performed and all variables which have a P value of less than 0.1 will be included in the multivariate analysis.




| | | Pradaxa<br>150mg | Pradaxa<br>(110 and 150 mg) |
|---|---|---|---|
| | Recovered with sequelae<br>Unknown<br>Fatal | | |
| Action Taken with Pradaxa (multi-response) | Dose not changed Dose reduced Dose increased Drug withdrawn | | |

Percentage calculated at patient level

Patients in the Safety Analysis Set. Subjects who receive at least one documented dose of study medication (Pradaxa®)

Table 55. Description of ADRs associated to BI product Pradaxa®

| | | Pradaxa<br>110mg | Pradaxa<br>150mg | Pradaxa<br>(110 and 150 mg) |
|---|---|---|---|---|
| ADRs associated to BI product (Pradaxa®) | Total ADRs | | | |
| Type of ADR | SOC1<br>PT11<br>PT12<br><br>SOC2<br>PT21<br>PT22 | | | |
| ADR outcome | Recovered Not yet recovered Recovered with sequelae Unknown Fatal | | | |
| Action Taken with Pradaxa | Dose not changed<br>Dose reduced<br>Dose increased<br>Drug withdrawn | | | |

Percentage calculated at event level

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to

<sup>.</sup> and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




Patients in the Safety Analysis Set. Subjects who receive at least one documented dose of study medication (Pradaxa®)

# 17.6 Serious Adverse Drug Reactions

Table 56. Patients with SADRs associated to BI product Pradaxa®

| | | Pradaxa<br>110mg | Pradaxa<br>150mg | Pradaxa<br>(110 and 150<br>mg) |
|---|---|---|---|---|
| SADRs associated to BI product | Total patients | | | |
| (Pradaxa®) | No | | | |
| | Yes | | | |
| Type of SADR | SOC1 | | | |
| (multi-response) | PT11 | | | |
| | PT12 | | | |
| | SOC2 | | | |
| | PT21 | | | |
| | PT22 | | | |
| Reason for seriousness | Results in death | | | |
| (multi-response) | Immediately life-threatening | | | |
| | Persistent or significant | | | |
| | disability/incapacity | | | |
| | Requires/prolongs hospitalization | | | |
| | Congenital anomaly/birth defect | | | |
| | Other comparable medical criteria | | | |
| SADR outcome | Recovered | | | |
| (multi-response) | Not yet recovered | | | |
| | Recovered with sequelae | | | |
| | Unknown | | | |
| | Fatal | | | |
| Action Taken with Pradaxa | Dose not changed | | | |
| (multi-response) | Dose reduced | | | |

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to




| | Pradaxa<br>(110 and 150<br>mg) |
|----------------------------------|--------------------------------|
| Dose increased<br>Drug withdrawn | |

Percentage calculated at patient level

Patients in the Safety Analysis Set. Subjects who receive at least one documented dose of study medication (Pradaxa®)

Table 57. Description of SADRs associated to BI product Pradaxa®

| | | Pradaxa<br>110mg | Pradaxa<br>150mg | Pradaxa<br>(110 and 150<br>mg) |
|---|---|---|---|---|
| SADRs associated to BI product (Pradaxa®) | Total SADRs | | | |
| Type of SADR | SOC1 | | | |
| (multi-response) | PT11 | | | |
| | PT12 | | | |
| | SOC2 | | | |
| | PT21 | | | |
| | PT22 | | | |
| Reason for seriousness | Results in death | | | |
| | Immediately life-threatening | | | |
| | Persistent or significant | | | |
| | disability/incapacity | | | |
| | Requires/prolongs hospitalization | | | |
| | Congenital anomaly/birth defect | | | |
| | Other comparable medical criteria | | | |
| SADR outcome | Recovered | | | |
| | Not yet recovered | | | |
| | Recovered with sequelae | | | |
| | Unknown | | | |
| | Fatal | | | |
| Action Taken with Pradaxa | Dose not changed | | | |
| | Dose reduced | | | |

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to

<sup>.</sup> and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




| | Pradaxa<br>150mg | Pradaxa<br>(110 and 150<br>mg) |
|---|---|---|
| Dose increased<br>Drug withdrawn | | |

Percentage calculated at event level

Patients in the Safety Analysis Set. Subjects who receive at least one documented dose of study medication (Pradaxa®)

# 17.7 Deaths

Table 58. List of deaths

| PATCOD | Adverse Event<br>Term | MedDRA<br>Code | Onset date | End date | Outcome | Relationship<br>with BI<br>product |
|---|---|---|---|---|---|---|

Document: H:\HOR-Europe\2019\2512352 - Study on anticoagulation management - BI\Proyecto\Estadistica\SAP\S

AP\_REBELD\_version1.0\_08072020.docx


Template No.: RWI TP BIOS0013 Revision 1 Reference: RWI WI BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to



| | | | a SECURE |
|---|---|---|---|
| Certificate Of Completion | | | |
| Envelope Id: D723D9040648460CA7C694EF256E<br>Subject: Please DocuSign: SAP_REBELD_version<br>Source Envelope: | | Status: Completed | |
| Document Pages: 108 Certificate Pages: 6 AutoNav: Enabled Envelopeld Stamping: Enabled Time Zone: (UTC+01:00) Amsterdam, Berlin, Berr | Signatures: 4 Initials: 0 n, Rome, Stockholm, Vienna | Envelope Originator: IP Address: | |
| Record Tracking | | | |
| Status: Original 7/10/2020 9:58:14 AM | Holder: | Location: DocuSign | |
| Signer Events | Signature | Timestamp | |
| | | Sent: 7/10/2020 10:04:50 AM<br>Viewed: 7/10/2020 10:51:57 A<br>Signed: 7/10/2020 10:55:25 Al | |
| Security Level: Email, Account Authentication (Required) | Signature Adoption: Pre-selected Style Signature ID: Using IP Address: With Signing Authentication via DocuSign password | | |
| Electronic Record and Signature Disclosure: Accepted: 7/10/2020 10:51:57 AM ID: | With Signing Reasons (on each tab): Soy el autor de este documento | | |
| Security Level: Email, Account Authentication (Required) | Signature Adoption: Pre-selected Style | Sent: 7/10/2020 10:55:36 AM<br>Resent: 7/13/2020 9:56:55 AM<br>Viewed: 7/13/2020 10:27:28 A<br>Signed: 7/13/2020 10:28:45 AM | M |
| | Signature ID: | | |

Using IP Address:

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab): He revisado este documento

Electronic Record and Signature Disclosure:
Accepted: 7/13/2020 10:27:28 AM
ID:

# **Signer Events** Signature **Timestamp** Sent: 7/13/2020 10:28:55 AM Viewed: 7/13/2020 11:04:08 AM Signed: 7/13/2020 11:05:15 AM Security Level: Email, Account Authentication Signature Adoption: Pre-selected Style (Required) Signature ID: Using IP Address: With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document **Electronic Record and Signature Disclosure:** Accepted: 6/16/2020 9:11:06 AM ID: Sent: 7/13/2020 11:05:24 AM Viewed: 7/13/2020 5:35:06 PM Signed: 7/13/2020 5:36:47 PM Security Level: Email, Account Authentication Signature Adoption: Pre-selected Style (Required) Signature ID: Using IP Address: With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I have reviewed this document **Electronic Record and Signature Disclosure:** Accepted: 7/10/2020 2:33:16 AM In Person Signer Events **Signature Timestamp Editor Delivery Events Status Timestamp Agent Delivery Events Status Timestamp Intermediary Delivery Events Status Timestamp Certified Delivery Events** Status Timestamp **Carbon Copy Events Status Timestamp** Sent: 7/13/2020 5:36:57 PM COPIED Validated Production Security Level: Email, Account Authentication (Required) **Electronic Record and Signature Disclosure:** Not Offered via DocuSign **Witness Events** Signature Timestamp **Notary Events** Signature **Timestamp**

**Timestamps** 

7/13/2020 5:36:57 PM

**Envelope Summary Events** 

**Envelope Sent** 

**Status** 

Hashed/Encrypted

| Envelope Summary Events | Status | Timestamps |
|---|---|---|
| Certified Delivered | Security Checked | 7/13/2020 5:36:57 PM |
| Signing Complete | Security Checked | 7/13/2020 5:36:57 PM |
| Completed | Security Checked | 7/13/2020 5:36:57 PM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Boehringer Ingelheim Validated Production (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

# Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

# Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

# Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

# **How to contact Boehringer Ingelheim Validated Production:**

| You may contact us to let us know of your changes as to how we may contact you electronic | onically. |
|---|---|
| to request paper copies of certain information from us, and to withdraw your prior conser | nt to |
| receive notices and disclosures electronically as follows: | |
| To contact us by email send messages to: | |
| <u> </u> | |

# To advise Boehringer Ingelheim Validated Production of your new email address

| To let us know of a change in your email address where we should send notices and disclosures |
|---|
| electronically to you, you must send an email message to us at |
| and in the body of such request you must state: your previous email address, your |
| new email address. We do not require any other information from you to change your email |
| address. |

If you created a DocuSign account, you may update it with your new email address through your account preferences.

#### To request paper copies from Boehringer Ingelheim Validated Production

| To request delivery from us of paper copies of the notices and disclosures previously provided |
|---|
| by us to you electronically, you must send us an email to |
| and in the body of such request you must state your email address, full name, |
| mailing address, and telephone number. We will bill you for any fees at that time, if any. |

# To withdraw your consent with Boehringer Ingelheim Validated Production

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

# Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

# Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Boehringer Ingelheim Validated Production as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Boehringer Ingelheim Validated Production during the course of your relationship with Boehringer Ingelheim Validated Production.